CLINICAL TRIAL: NCT00985673
Title: A Study to Evaluate the Safety and Immunogenicity of an A/California/7/2009 (H1N1)V-like Vaccine GSK2340274A or GSK2340273A Co-administered With Trivalent Inactivated Seasonal Influenza Vaccine in Adults 19 to 40 Years of Age
Brief Title: Safety and Immunogenicity of H1N1 Vaccine With Trivalent Inactivated Seasonal Influenza Vaccine in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 113536
Record Dates: First submitted 2009-09-24; First posted 2009-09-28 (Estimated); Results first posted 2012-01-30 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2016-09

CONDITIONS: Influenza
Keywords: GSK Bio's influenza vaccine GSK2340274A; influenza infection; GSK Bio's influenza vaccine GSK2340273A
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (6):
- Flulaval/placebo/unadjuvanted Arepanrix Group (Experimental): subjects received co-administration of Flulaval vaccine and saline placebo on Day 0 followed by the unadjuvanted formulation of Arepanrix vaccine on Day 21 and Day 42. All vaccines were administered intramuscularly in the deltoids of the dominant or non dominant arm. At Day 0 the two vaccines were administered each in a separate arm, at Day 21 in the dominant arm and at Day 42 in the non-dominant arm.
  Interventions: Biological: GSK2340273A; Biological: Seasonal trivalent influenza vaccine (TIV); Biological: Saline placebo
- Flulaval/placebo/Arepanrix Group (Experimental): subjects received co-administration of Flulaval vaccine and saline placebo on Day 0 followed the administration of Arepanrix vaccine on Day 21 and Day 42. All vaccines were administered intramuscularly in the deltoids of the dominant or non dominant arm. At Day 0 the two vaccines were administered each in a separate arm, at Day 21 in the dominant arm and at Day 42 in the non-dominant arm.
  Interventions: Biological: GSK2340274A; Biological: Seasonal trivalent influenza vaccine (TIV); Biological: Saline placebo
- Flulaval/unadjuvanted Arepanrix/placebo Group (Experimental): subjects received co-administration of Flulaval vaccine and the unadjuvanted formulation of Arepanrix vaccine on Day 0 followed by the administration of the unadjuvanted formulation of Arepanrix vaccine on Day 21 and saline placebo on Day 42. All vaccines were administered intramuscularly in the deltoids of the dominant or non dominant arm. At Day 0 the two vaccines were administered each in a separate arm, at Day 21 in the dominant arm and at Day 42 in the non-dominant arm.
  Interventions: Biological: GSK2340273A; Biological: Seasonal trivalent influenza vaccine (TIV); Biological: Saline placebo
- Flulaval/Arepanrix/placebo Group (Experimental): subjects received co-administration of Flulaval vaccine and Arepanrix vaccine on Day 0 followed by Arepanrix vaccine on Day 21 and saline placebo on Day 42. All vaccines were administered intramuscularly in the deltoids of the dominant or non dominant arm. At Day 0 the two vaccines were administered each in a separate arm, at Day 21 in the dominant arm and at Day 42 in the non-dominant arm.
  Interventions: Biological: GSK2340274A; Biological: Seasonal trivalent influenza vaccine (TIV); Biological: Saline placebo
- Unadjuvanted Arepanrix/placebo/Flulaval Group (Experimental): subjects received co-administration of the unadjuvanted formulation of Arepanrix vaccine and saline placebo on Day 0 followed by the unadjuvanted formulation of Arepanrix vaccine on Day 21 and Flulaval vaccine on Day 42. All vaccines were administered intramuscularly in the deltoids of the dominant or non dominant arm. At Day 0 the two vaccines were administered each in a separate arm, at Day 21 in the dominant arm and at Day 42 in the non-dominant arm.
  Interventions: Biological: GSK2340273A; Biological: Seasonal trivalent influenza vaccine (TIV); Biological: Saline placebo
- Arepanrix/placebo/Flulaval Group (Experimental): subjects received co-administration of Arepanrix vaccine and saline placebo on Day 0 followed by Arepanrix vaccine on Day 21 and Flulaval vaccine on Day 42. All vaccines were administered intramuscularly in the deltoids of the dominant or non dominant arm. At Day 0 the two vaccines were administered each in a separate arm, at Day 21 in the dominant arm and at Day 42 in the non-dominant arm.
  Interventions: Biological: GSK2340274A; Biological: Seasonal trivalent influenza vaccine (TIV); Biological: Saline placebo

INTERVENTIONS:
Biological: GSK2340274A — Two intramuscular injections
  Arms: Arepanrix/placebo/Flulaval Group; Flulaval/Arepanrix/placebo Group; Flulaval/placebo/Arepanrix Group
Biological: GSK2340273A — Two intramuscular injections
  Arms: Flulaval/placebo/unadjuvanted Arepanrix Group; Flulaval/unadjuvanted Arepanrix/placebo Group; Unadjuvanted Arepanrix/placebo/Flulaval Group
Biological: Seasonal trivalent influenza vaccine (TIV) — Single intramuscular injection
Biological: Saline placebo — Single intramuscular injection

SUMMARY:
The purpose of this study is to characterize the safety and immunogenicity of the H1N1 (swine) flu vaccines GSK2340274A and GSK2340273A when co-administered with the seasonal flu vaccine in adults 19 to 40 years of age.

DETAILED DESCRIPTION:
Collaborators: United States Department of Health and Human Services, Office of Biomedical Advanced Research and Development Authority

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject.
* Male or female adults, 19-40 years of age at the time of the first vaccination.
* Safety laboratory tests results within the parameters specified in the protocol.
* Satisfactory baseline medical assessment by physical examination.
* Comprehension of the study requirements, ability to comprehend and comply with procedures for collection of safety data, expressed availability for the required study period, and ability and willingness to attend scheduled visits as documented by signature on the informed consent document.
* Access to a consistent means of telephone contact, which may be either in the home or at the workplace, land line, or mobile, but NOT a pay phone or other multiple-user device.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:
* has practiced adequate contraception for 30 days prior to vaccination, and
* has a negative pregnancy test on the day of first vaccination, and
* has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Previous vaccination with an H1N1v-like virus vaccine or a medical history of physician-confirmed infection with an H1N1v-like virus.
* Prior receipt at any time of any seasonal influenza vaccine.
* Planned administration of any vaccine not foreseen by the study protocol between Day 0 and the Day 63 phlebotomy.
* Administration of any licensed vaccine within 4 weeks before the first study vaccine dose.
* Use of any investigational or non-registered product other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Receipt of systemic glucocorticoids within one month prior to study enrolment, or any other cytotoxic or immunosuppressive drug within six months of study enrolment. Topical, intra-articularly injected, or inhaled glucocorticoids, topical calcineurin inhibitors or imiquimod are allowed.
* Receipt of any immunoglobulins and/or any blood products within three months of study enrolment or planned administration of any of these products during the study period.
* Presence of evidence of substance abuse or of neurological or psychiatric diagnoses which, even if stable, are deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Presence of a temperature >= 38.0ºC (>=100.4ºF), or acute symptoms greater than "mild" severity on the scheduled date of first vaccination.
* Diagnosed with cancer, or treatment for cancer, within 3 years.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Any significant disorder of coagulation or treatment with warfarin derivatives or heparin. Persons receiving individual doses of low molecular weight heparin outside of 24 hours prior to vaccination are eligible. Persons receiving prophylactic antiplatelet medications, e.g., low-dose acetylsalicylic acid, and without a clinically-apparent bleeding tendency, are eligible.
* An acute evolving neurological disorder or history of Guillain-Barré syndrome within six weeks of receipt of seasonal influenza vaccine.
* Any known or suspected allergy to any constituent of influenza vaccines; a history of anaphylactic-type reaction to any constituent of influenza vaccines; or a history of severe adverse reaction to a previous influenza vaccine.
* Known pregnancy or a positive urine beta-human chorionic gonadotropin test result prior to first vaccination.
* Lactating or nursing women.

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 611 (Actual)
Dates: Start 2009-10-01; Primary Completion 2009-12-28 (Actual); Study Completion 2010-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- United States (4):
  - GSK Investigational Site, Stockbridge, Georgia
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Fort Worth, Texas
- Canada (3):
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Friel D, Co M, Ollinger T, Salaun B, Schuind A, Li P, Walravens K, Ennis FA, Vaughn DW. Non-neutralizing antibody responses following A(H1N1)pdm09 influenza vaccination with or without AS03 adjuvant system. Influenza Other Respir Viruses. 2021 Jan;15(1):110-120. doi: 10.1111/irv.12780. Epub 2020 Sep 5. PMID 32889792
- [Derived] Langley JM, Frenette L, Chu L, McNeil S, Halperin S, Li P, Vaughn D. A randomized, controlled non-inferiority trial comparing A(H1N1)pmd09 vaccine antigen, with and without AS03 adjuvant system, co-administered or sequentially administered with an inactivated trivalent seasonal influenza vaccine. BMC Infect Dis. 2012 Oct 30;12:279. doi: 10.1186/1471-2334-12-279. PMID 23110320
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 113536 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113536 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113536 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113536 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113536 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113536 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113536 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Started | 102 | 104 | 102 | 100 | 101 | 102
Completed | 95 | 93 | 90 | 88 | 93 | 96
Not Completed | 7 | 11 | 12 | 12 | 8 | 6
Not completed — Lost to Follow-up | 6 | 7 | 6 | 10 | 5 | 3
Not completed — Withdrawal by Subject | 0 | 4 | 5 | 2 | 2 | 3
Not completed — Other | 1 | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group | Total
Number analyzed (Participants) | 102 | 104 | 102 | 100 | 101 | 102 | 611
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.7 (6.20) | 28.6 (6.24) | 28.2 (6.32) | 29.2 (6.12) | 29.3 (6.47) | 28.1 (6.08) | 28.9 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 62 | 54 | 48 | 60 | 58 | 335
  Male | 49 | 42 | 48 | 52 | 41 | 44 | 276

OUTCOME MEASURES:

1. Primary Outcome: Hemagglutination Inhibition (HI) Antibody Titers Against A/California/7/2009 H1N1 Vaccine Strain.
Description: The A/California vaccine virus-homologous antibody response was measured in subjects having received Flulaval vaccine co-administered with the first dose of Arepanrix vaccine, and in subjects having received two doses of Arepanrix vaccine alone.
  Titers were expressed as geometric mean antibody titers (GMTs).
Time Frame: 21 days after the second dose of Arepanrix vaccine (at Day 42).
Population: The According-To-Protocol (ATP) cohort for immunogenicity included evaluable subjects (i.e. those meeting eligibility criteria, with no elimination criteria) who received 2 doses and for whom assay results were available for antibodies against H1N1 antigen 21 days after the 2nd vaccine dose.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Number analyzed (Participants) | 0 | 0 | 0 | 89 | 0 | 91
Titers |  |  |  | 589.8 [517.8 to 671.8] |  | 933.1 [815.6 to 1067.6]

2. Primary Outcome: Hemagglutination Inhibition (HI) Antibody Titers Against A/California/7/2009 H1N1 Vaccine Strain.
Description: The A/California vaccine virus-homologous antibody response was measured in subjects having received Flulaval vaccine co-administered with the first dose of the unadjuvanted formulation of Arepanrix vaccine, and in subjects having received two doses of the unadjuvanted formulation of Arepanrix vaccine alone.
  Titers were expressed as geometric mean antibody titers (GMTs).
Time Frame: 21 days after the second dose of the unadjuvanted formulation of Arepanrix vaccine (at Day 42)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Number analyzed (Participants) | 0 | 0 | 92 | 0 | 91 | 0
Titers |  |  | 271.2 [224.6 to 327.4] |  | 387.1 [314.4 to 476.7] |

3. Secondary Outcome: Number of Influenza-specific Cluster of Differentiation 4 (CD4) T-cells Per Million Producing Two or More Markers Within Cluster Differentiation 40 Ligand (CD40L), Interleukin-2 (IL-2), Interferon-γ (IFN-γ) and Tumor Necrosis Factor-α (TNF-α).
Description: Influenza-specific CD4 T-Cells were stimulated in vitro with A/California virus and seasonal Influenza viruses, related antigens or derived peptides.
  Stimulating antigens were A/Brisbane, A/California, pool peptides H1N1 and pool FLU.
Time Frame: On Days 0, 7, 21, 28, 42, 63 and 182
Population: The According-To-Protocol (ATP) cohort for immunogenicity at Day 182 included evaluable subjects (i.e. those meeting eligibility criteria, with no elimination criteria) for whom 1 dose of Flulaval vaccine and 2 doses of pandemic vaccine were administered and results were available for antibodies against H1N1 antigen at day 182.
Measure: Mean (Standard Deviation); unit: Number of T cells/million
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 25 | 28
Number of T cells/million
  A/Brisbane [D0] (N=25,25,24,25,25,26) | 2533.40 (1225.90) | 2604.64 (1435.48) | 3521.33 (1922.24) | 2612.56 (1256.47) | 2644.40 (1219.04) | 2016.31 (822.34)
  A/Brisbane [D7] (N=24,27,24,23,24,26) | 4437.33 (1930.30) | 4595.26 (2058.76) | 5560.33 (3301.90) | 6242.30 (2773.60) | 4269.96 (1744.37) | 4674.88 (2325.77)
  A/Brisbane [D21] (N=26,25,27,24,24,26) | 3561.00 (1502.24) | 3756.72 (1379.69) | 5581.78 (3123.38) | 6069.67 (3306.79) | 3894.54 (1596.44) | 5590.23 (2407.32)
  A/Brisbane [D28] (N=27,27,27,26,25,27) | 3500.22 (1615.89) | 4269.11 (1482.01) | 5102.78 (2856.77) | 6989.15 (3950.45) | 3816.20 (1290.25) | 7083.19 (3227.04)
  A/Brisbane [D42] (N=27,26,27,27,24,28) | 3595.11 (1268.17) | 5246.88 (2407.94) | 4791.41 (2706.43) | 5607.96 (2773.17) | 3872.67 (1270.26) | 6200.64 (2733.75)
  A/Brisbane [D63] (N=26,26,25,25,24,26) | 3407.62 (1114.62) | 6444.50 (2681.50) | 4169.32 (2216.49) | 5020.88 (2346.39) | 4074.38 (1639.45) | 5757.04 (3131.86)
  A/Brisbane [D182] (N=26,24,26,26,25,25) | 3190.31 (1086.38) | 4631.00 (1834.57) | 4132.81 (1816.70) | 3988.04 (1606.16) | 3672.16 (1191.85) | 4568.16 (2043.61)
  A/California [D0] (N=25,25,24,25,25,26) | 2176.28 (1226.08) | 1988.24 (1072.73) | 2804.63 (1912.94) | 2055.44 (1053.95) | 2109.52 (828.11) | 1641.04 (799.39)
  A/California [D7] (N=24,27,24,23,24,26) | 4089.25 (2131.69) | 3852.44 (1970.35) | 4780.21 (2828.25) | 5265.74 (2008.41) | 3224.42 (1238.08) | 3590.08 (1912.94)
  A/California [D21] (N=26,25,27,24,24,26) | 3144.62 (1723.51) | 3032.52 (1342.30) | 4455.00 (2768.12) | 4986.71 (2398.42) | 2975.38 (1058.31) | 4793.35 (2194.74)
  A/California [D28] (N=27,27,27,26,25,27) | 3061.63 (1632.58) | 3770.44 (1460.62) | 4058.63 (2349.19) | 5979.12 (3448.84) | 2875.52 (837.73) | 6689.44 (3501.59)
  A/California [D42] (N=27,27,27,27,24,28) | 2931.04 (1276.42) | 4381.48 (2053.51) | 3720.07 (2261.08) | 4658.07 (1939.82) | 2838.00 (1008.20) | 5622.14 (2870.26)
  A/California [D63] (N=26,26,25,25,24,26) | 2768.15 (1109.96) | 5328.19 (2436.59) | 3149.00 (1844.25) | 3967.12 (1655.09) | 3246.71 (1379.49) | 5151.62 (3008.33)
  A/California [D182] (N=26,24,26,26,25,25) | 1461.88 (735.77) | 2333.88 (925.38) | 1838.96 (842.26) | 2068.73 (939.92) | 1630.40 (592.23) | 2513.48 (1232.20)
  Pool peptides H1 [D0] (N=25,24,24,25,23,25) | 349.64 (336.13) | 428.00 (296.76) | 356.79 (206.44) | 320.52 (216.19) | 443.35 (356.02) | 271.76 (180.44)
  Pool peptides H1 [D7] (N=24,27,24,23,24,25) | 596.42 (500.15) | 581.63 (527.07) | 708.96 (518.87) | 857.04 (474.48) | 692.29 (454.48) | 718.76 (663.81)
  Pool peptides H1 [D21] (N=26,24,27,24,24,26) | 465.42 (352.18) | 589.79 (459.57) | 728.15 (623.89) | 974.67 (579.23) | 619.50 (391.47) | 1022.38 (572.50)
  Pool peptides H1 [D28] (N=26,27,27,26,25,27) | 480.42 (392.81) | 704.59 (518.63) | 528.78 (322.10) | 1345.69 (1536.94) | 642.00 (379.90) | 1251.07 (695.04)
  Pool peptides H1 [D42] (N=27,27,27,27,24,28) | 467.70 (302.91) | 1049.96 (865.58) | 514.78 (296.67) | 1080.93 (669.26) | 600.04 (496.71) | 1228.25 (637.35)
  Pool peptides H1 [D63] (N=26,26,25,25,24,26) | 504.92 (321.17) | 1248.54 (1175.35) | 460.28 (267.85) | 815.24 (634.45) | 508.58 (316.75) | 910.81 (482.86)
  Pool peptides H1 [D182] (N=26,24,26,26,25,25) | 554.65 (439.30) | 824.17 (565.53) | 531.73 (481.91) | 648.69 (557.34) | 552.52 (528.46) | 757.68 (638.40)
  Pool Flu [D0] (N=24,25,24,25,25,24) | 3286.63 (1710.00) | 3531.36 (1972.37) | 4315.71 (2499.77) | 3056.80 (1096.38) | 3308.08 (1124.49) | 2775.50 (1214.18)
  Pool Flu [D7] (N=24,27,24,23,24,25) | 6574.50 (3399.35) | 6921.85 (4366.14) | 7096.46 (3777.79) | 7682.43 (2951.47) | 4668.17 (1675.47) | 4713.28 (2161.14)
  Pool Flu [D21] (N=25,25,27,24,24,25) | 5234.16 (2513.78) | 5124.60 (2268.53) | 6579.26 (3489.20) | 6949.96 (3006.25) | 4329.96 (1672.20) | 5691.08 (2047.10)
  Pool Flu [D28] (N=25,27,27,26,25,26) | 4767.36 (2217.82) | 5256.07 (2292.16) | 6090.00 (3336.49) | 7265.23 (3520.63) | 4047.92 (1219.00) | 6804.42 (2824.80)
  Pool Flu [D42] (N=26,27,27,26,24,27) | 4734.42 (1823.28) | 5881.78 (2641.14) | 5721.70 (3058.63) | 6239.38 (2542.17) | 4167.63 (1351.74) | 6215.93 (2389.59)
  Pool Flu [D63] (N=25,26,25,25,24,24) | 4405.96 (1586.42) | 6639.92 (3131.66) | 4893.88 (2322.10) | 5323.84 (2132.52) | 4900.17 (2016.61) | 6455.25 (2694.48)
  Pool Flu [D182] (N=26,24,26,26,25,25) | 3304.50 (1393.44) | 4325.63 (1541.34) | 4006.46 (1836.30) | 3937.67 (1413.94) | 3918.28 (1284.32) | 4277.76 (1655.16)

4. Secondary Outcome: Number of Influenza-specific Cluster of Differentiation 8 (CD8) T-cells Per Million Producing Two or More Markers Within Cluster Differentiation 40 Ligand (CD40L), Interleukin-2 (IL-2), Interferon-γ (IFN-γ) and Tumor Necrosis Factor-α (TNF-α).
Description: Influenza-specific CD8 T-Cells were stimulated in vitro with A/California virus and seasonal Influenza viruses, related antigens or derived peptides.
  Stimulating antigens were A/Brisbane, A/California, pool peptides H1N1 and pool FLU.
Time Frame: On Days 0, 7, 21, 28, 42, 63 and 182
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Number of T cells/million
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 25 | 28
Number of T cells/million
  A/Brisbane [D0] (N=25,25,24,25,25,26) | 515.36 (1191.10) | 382.84 (595.58) | 489.08 (520.30) | 183.96 (226.54) | 1222.40 (4485.04) | 119.46 (113.79)
  A/Brisbane [D7] (N=24,27,24,23,24,26) | 772.96 (716.40) | 884.81 (1225.90) | 1115.96 (1545.07) | 725.39 (585.98) | 1611.96 (4894.45) | 529.73 (416.76)
  A/Brisbane [D21] (N=26,25,27,24,24,26) | 601.31 (1154.73) | 517.44 (799.20) | 655.22 (1327.00) | 319.17 (315.86) | 1184.17 (4146.13) | 501.08 (1319.91)
  A/Brisbane [D28] (N=27,27,27,26,25,27) | 629.22 (964.11) | 642.22 (850.79) | 498.33 (730.34) | 508.88 (540.73) | 1466.76 (5768.96) | 1735.48 (5219.43)
  A/Brisbane [D42] (N=27,26,27,27,24,28) | 666.67 (1180.05) | 551.88 (911.02) | 525.07 (938.18) | 209.07 (171.21) | 1737.50 (6861.67) | 501.54 (1329.90)
  A/Brisbane [D63] (N=26,26,25,25,24,26) | 620.00 (1393.77) | 420.50 (486.62) | 428.92 (687.17) | 230.84 (226.10) | 1493.46 (5828.76) | 529.81 (1383.73)
  A/Brisbane [D182] (N=26,24,26,26,25,25) | 550.27 (1948.06) | 436.79 (653.50) | 377.65 (426.59) | 86.81 (99.38) | 1474.56 (6012.19) | 370.64 (955.57)
  A/California [D0] (N=25,25,24,25,25,26) | 357.40 (800.46) | 189.28 (197.92) | 271.58 (192.68) | 365.72 (985.87) | 482.64 (1286.27) | 93.50 (114.90)
  A/California [D7] (N=24,27,24,23,24,26) | 610.29 (744.70) | 466.93 (573.69) | 716.88 (1251.20) | 553.78 (639.15) | 834.50 (2063.34) | 348.69 (326.74)
  A/California [D21] (N=26,25,27,24,24,26) | 332.00 (539.48) | 275.04 (334.83) | 324.37 (668.77) | 183.00 (146.43) | 428.92 (1071.57) | 351.69 (713.52)
  A/California [D28] (N=27,27,27,26,25,27) | 470.33 (655.02) | 452.93 (547.61) | 332.63 (553.07) | 344.54 (288.96) | 973.96 (3644.93) | 497.67 (612.95)
  A/California [D42] (N=27,27,27,27,24,28) | 314.89 (289.95) | 304.00 (255.38) | 247.89 (459.58) | 157.67 (192.15) | 702.50 (2209.62) | 291.96 (654.16)
  A/California [D63] (N=26,2625,25,24,26) | 203.62 (197.89) | 260.54 (359.88) | 242.36 (357.21) | 114.24 (165.15) | 853.83 (3236.11) | 194.73 (453.09)
  A/California [D182] (N=26,24,26,26,25,25) | 214.85 (326.43) | 220.71 (330.88) | 225.50 (366.51) | 139.50 (273.43) | 598.92 (2344.64) | 138.52 (245.14)
  Pool peptides H1 [D0] (N=25,24,24,25,23,25) | 110.48 (140.31) | 180.38 (359.58) | 101.04 (158.31) | 150.08 (215.56) | 111.26 (162.75) | 70.92 (113.24)
  Pool peptides H1 [D7] (N=24,27,24,23,24,25) | 205.33 (288.67) | 185.15 (243.88) | 202.13 (293.11) | 254.65 (417.53) | 243.46 (382.39) | 173.48 (202.67)
  Pool peptides H1 [D21] (N=26,24,27,24,24,26) | 103.81 (160.76) | 194.92 (384.18) | 101.30 (148.62) | 140.75 (155.63) | 211.96 (482.54) | 173.77 (432.74)
  Pool peptides H1 [D28] (N=26,27,27,26,25,27) | 100.08 (132.13) | 170.04 (385.99) | 124.56 (181.86) | 277.77 (329.71) | 160.80 (216.87) | 187.37 (361.53)
  Pool peptides H1 [D42] (N=27,27,27,27,24,28) | 143.67 (189.28) | 157.41 (350.83) | 87.41 (115.12) | 103.89 (139.95) | 266.75 (481.50) | 145.96 (261.67)
  Pool peptides H1 [D63] (N=26,26,25,25,24,26) | 85.96 (97.66) | 173.88 (244.91) | 113.20 (193.78) | 88.28 (162.10) | 210.33 (403.19) | 88.19 (206.24)
  Pool peptides H1 [D182] (N=26,24,26,26,25,25) | 287.31 (511.19) | 265.63 (343.36) | 306.04 (630.16) | 241.42 (353.02) | 255.44 (425.71) | 198.44 (561.99)
  Pool Flu [D0] (N=24,25,24,25,25,24) | 351.38 (467.93) | 224.60 (251.59) | 478.42 (463.43) | 344.60 (641.98) | 761.68 (2411.00) | 157.63 (166.45)
  Pool Flu [D7] (N=24,27,24,23,24,25) | 986.92 (863.16) | 843.44 (826.65) | 1042.17 (1237.44) | 788.78 (947.53) | 1094.96 (3111.41) | 522.84 (514.35)
  Pool Flu [D21] (N=25,25,27,24,24,25) | 586.32 (876.08) | 268.24 (324.48) | 609.07 (997.10) | 266.63 (252.28) | 693.88 (2082.82) | 406.28 (620.10)
  Pool Flu [D28] (N=25,27,27,26,25,26) | 484.48 (587.46) | 508.11 (559.97) | 505.33 (595.15) | 458.12 (496.69) | 963.20 (3548.16) | 423.62 (430.29)
  Pool Flu [D42] (N=26,27,27,26,24,27) | 506.35 (560.83) | 356.41 (392.23) | 471.30 (610.38) | 344.77 (709.66) | 996.67 (3648.68) | 391.11 (755.53)
  Pool Flu [D63] (N=25,26,25,25,24,24) | 461.20 (698.48) | 325.12 (270.84) | 402.24 (418.89) | 296.08 (624.75) | 1123.13 (4008.27) | 432.08 (1145.71)
  Pool Flu [D182] (N=26,24,26,26,25,25) | 404.77 (981.01) | 315.75 (441.50) | 334.23 (447.12) | 291.73 (790.15) | 926.40 (3463.27) | 234.92 (398.06)

5. Secondary Outcome: Number of Subjects Reporting Clinical Laboratory Abnormalities in Biochemical and Haematological Parameters Assessed
Description: Laboratory parameters assessed were alanine aminotransferase (ALAT), aspartate aminotransferase (ASAT), alkaline phosphatase (AP), bilirubin (BIL) (total (T)), basophils (BAS). For each parameter and for each range it was assessed whether the values of the subjects were in unkown, above, below or within the range.
Time Frame: On Days 0, 7, 21, 28, 42, 63 and 182
Population: The Total Vaccinated Cohort included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Number analyzed (Participants) | 102 | 104 | 102 | 100 | 101 | 102
Subjects
  ALAT [D0] Below (N=102,101,102,100,101,102) | 0 | 0 | 0 | 0 | 0 | 0
  ALAT [D0] Within (N=102,101,102,100,101,102) | 100 | 101 | 99 | 95 | 100 | 99
  ALAT [D0] Above (N=102,101,102,100,101,102) | 2 | 3 | 2 | 4 | 0 | 3
  ALAT [D7] Below (N=102,101,100,99,100,99) | 0 | 0 | 0 | 0 | 0 | 0
  ALAT [D7] Within (N=102,101,100,99,100,99) | 100 | 96 | 99 | 97 | 100 | 98
  ALAT [D7] Above (N=102,101,100,99,100,99) | 2 | 5 | 1 | 2 | 0 | 1
  ALAT [D21] Below (N=101,100,97,97,99,99) | 0 | 0 | 0 | 0 | 0 | 0
  ALAT [D21] Within (N=101,100,97,97,99,99) | 96 | 97 | 96 | 96 | 96 | 97
  ALAT [D21] Above (N=101,100,97,97,99,99) | 5 | 3 | 1 | 1 | 3 | 1
  ALAT [D28] Below (N=101,98,96,98,98,97) | 0 | 0 | 0 | 0 | 0 | 0
  ALAT [D28] Within (N=101,98,96,98,98,97) | 96 | 96 | 94 | 93 | 96 | 92
  ALAT [D28] Above (N=101,98,96,98,98,97) | 4 | 2 | 2 | 4 | 2 | 4
  ALAT [D42] Below (N=101,97,95,95,96,97) | 0 | 0 | 0 | 0 | 0 | 0
  ALAT [D42] Within (N=101,97,95,95,96,97) | 97 | 94 | 93 | 94 | 92 | 95
  ALAT [D42] Above (N=101,97,95,95,96,97) | 4 | 3 | 1 | 1 | 2 | 2
  ALAT [D63] Below (N=100,95,95,95,97,97) | 0 | 0 | 0 | 0 | 0 | 0
  ALAT [D63] Within (N=100,95,95,95,97,97) | 93 | 89 | 93 | 95 | 93 | 92
  ALAT [D63] Above (N=100,95,95,95,97,97) | 6 | 5 | 1 | 0 | 3 | 3
  ALAT [D182] Below (N=99,91,88,91,93,97) | 0 | 0 | 0 | 0 | 0 | 0
  ALAT [D182] Within (N=99,91,88,91,93,97) | 97 | 89 | 88 | 90 | 91 | 95
  ALAT [D182] Above (N=99,91,88,91,93,97) | 2 | 1 | 0 | 1 | 1 | 2
  AP [D0] Below (N=102,104, 102,100,101,102) | 0 | 0 | 0 | 0 | 0 | 0
  AP [D0] Within (N=102,104, 102,100,101,102) | 102 | 104 | 100 | 98 | 99 | 101
  AP [D0] Above (N=102,104, 102,100,101,102) | 0 | 0 | 1 | 1 | 1 | 1
  AP [D7] Below (N=102,101,100,99,100,99) | 0 | 0 | 0 | 0 | 0 | 0
  AP [D7] Within (N=102,101,100,99,100,99) | 101 | 101 | 100 | 98 | 99 | 98
  AP [D7] Above (N=102,101,100,99,100,99) | 1 | 0 | 0 | 1 | 1 | 1
  AP [D21] Below (N=101,100,97,97,99,99) | 0 | 0 | 0 | 0 | 0 | 0
  AP [D21] Within (N=101,100,97,97,99,99) | 101 | 100 | 96 | 96 | 97 | 97
  AP [D21] Above (N=101,100,97,97,99,99) | 0 | 0 | 1 | 1 | 2 | 1
  AP [D28] Below (N=101,98,96,98,98,97) | 0 | 0 | 0 | 0 | 0 | 0
  AP [D28] Within (N=101,98,96,98,98,97) | 99 | 97 | 95 | 95 | 98 | 96
  AP [D28] Above (N=101,98,96,98,98,97) | 1 | 1 | 1 | 2 | 0 | 0
  AP [D42] Below (N=101,97, 95,95,96,97) | 0 | 0 | 0 | 0 | 0 | 0
  AP [D42] Within (N=101,97, 95,95,96,97) | 99 | 97 | 94 | 92 | 93 | 96
  AP [D42] Above (N=101,97, 95,95,96,97) | 2 | 0 | 0 | 3 | 1 | 1
  AP [D63] Below (N=100,95,95,95,97,97) | 0 | 0 | 0 | 0 | 0 | 0
  AP [D63] Within (N=100,95,95,95,97,97) | 99 | 94 | 93 | 92 | 95 | 94
  AP [D63] Above (N=100,95,95,95,97,97) | 0 | 0 | 1 | 3 | 1 | 1
  AP [D182] Below (N=99,91,88,91,93,97) | 0 | 0 | 0 | 0 | 0 | 0
  AP [D182] Within (N=99,91,88,91,93,97) | 98 | 90 | 88 | 90 | 89 | 97
  AP [D182] Above (N=99,91,88,91,93,97) | 1 | 0 | 0 | 1 | 3 | 0
  ASAT [D0] Below (N=102,104,102,100,101,102) | 0 | 0 | 0 | 0 | 0 | 0
  ASAT [D0] Within (N=102,104,102,100,101,102) | 101 | 102 | 100 | 98 | 99 | 101
  ASAT [D0] Above (N=102,104,102,100,101,102) | 1 | 2 | 1 | 1 | 1 | 1
  ASAT [D7] Below (N=102,101,100,99,100,99) | 0 | 0 | 0 | 0 | 0 | 0
  ASAT [D7] Within (N=102,101,100,99,100,99) | 99 | 99 | 97 | 99 | 99 | 97
  ASAT [D7] Above (N=102,101,100,99,100,99) | 3 | 2 | 2 | 0 | 1 | 2
  ASAT [D21] Below (N=101,100,97,97,99,99) | 0 | 0 | 0 | 0 | 0 | 0
  ASAT [D21] Within (N=101,100,97,97,99,99) | 99 | 99 | 97 | 97 | 98 | 97
  ASAT [D21] Above (N=101,100,97,97,99,99) | 2 | 1 | 0 | 0 | 1 | 1
  ASAT [D28] Below (N=101,98,96,98,98,97) | 0 | 0 | 0 | 0 | 0 | 0
  ASAT [D28] Within (N=101,98,96,98,98,97) | 96 | 97 | 93 | 95 | 98 | 93
  ASAT [D28] Above (N=101,98,96,98,98,97) | 4 | 1 | 3 | 2 | 0 | 3
  ASAT [D42] Below (N=101,97,95,95,96,97) | 0 | 0 | 0 | 0 | 0 | 0
  ASAT [D42] Within (N=101,97,95,95,96,97) | 95 | 95 | 93 | 95 | 94 | 97
  ASAT [D42] Above (N=101,97,95,95,96,97) | 6 | 2 | 1 | 0 | 0 | 0
  ASAT [D63] Below (N=100,95,95,95,97,97) | 0 | 0 | 0 | 0 | 0 | 0
  ASAT [D63] Within (N=100,95,95,95,97,97) | 98 | 94 | 92 | 94 | 95 | 93
  ASAT [D63] Above (N=100,95,95,95,97,97) | 1 | 0 | 1 | 1 | 0 | 2
  ASAT [D182] Below (N=99,91,88,91,93,97) | 0 | 0 | 0 | 0 | 0 | 0
  ASAT [D182] Within (N=99,91,88,91,93,97) | 96 | 86 | 87 | 88 | 91 | 97
  ASAT [D182] Above (N=99,91,88,91,93,97) | 2 | 4 | 0 | 3 | 1 | 0
  BAS [D0] Below (N=102,104,102,100,101,102) | 0 | 0 | 0 | 0 | 0 | 0
  BAS [D0] Within (N=102,104,102,100,101,102) | 100 | 104 | 102 | 98 | 101 | 102
  BAS [D0] Above (N=102,104,102,100,101,102) | 0 | 0 | 0 | 0 | 0 | 0
  BAS [D7] Below (N=102,101,100,99,100,99) | 0 | 0 | 0 | 0 | 0 | 0
  BAS [D7] Within (N=102,101,100,99,100,99) | 102 | 100 | 100 | 98 | 100 | 99
  BAS [D7] Above (N=102,101,100,99,100,99) | 0 | 0 | 0 | 0 | 0 | 0
  BAS [D21] Below (N=101,100,97,97,99,99) | 0 | 0 | 0 | 0 | 0 | 0
  BAS [D21] Within (N=101,100,97,97,99,99) | 101 | 99 | 94 | 96 | 97 | 95
  BAS [D21] Above (N=101,100,97,97,99,99) | 0 | 0 | 0 | 0 | 0 | 0
  BAS [D28] Below (N=101,98,96,98,98,97) | 0 | 0 | 0 | 0 | 0 | 0
  BAS [D28] Within (N=101,98,96,98,98,97) | 99 | 96 | 96 | 96 | 97 | 94
  BAS [D28] Above (N=101,98,96,98,98,97) | 0 | 0 | 0 | 0 | 0 | 0
  BAS [D42] Below (N=101,97,95,95,96,97) | 0 | 0 | 0 | 0 | 0 | 0
  BAS [D42] Within (N=101,97,95,95,96,97) | 101 | 97 | 95 | 95 | 96 | 97
  BAS [D42] Above (N=101,97,95,95,96,97) | 0 | 0 | 0 | 0 | 0 | 0
  BAS [D63] Below (N=100,95,95,95,97,97) | 0 | 0 | 0 | 0 | 0 | 0
  BAS [D63] Within (N=100,95,95,95,97,97) | 100 | 95 | 95 | 95 | 97 | 97
  BAS [D63] Above (N=100,95,95,95,97,97) | 0 | 0 | 0 | 0 | 0 | 0
  BAS [D182] Below (N=99,91,88,91,93,97) | 0 | 0 | 0 | 0 | 0 | 0
  BAS [D182] Within (N=99,91,88,91,93,97) | 99 | 91 | 88 | 89 | 93 | 96
  BAS [D182] Above (N=99,91,88,91,93,97) | 0 | 0 | 0 | 0 | 0 | 0
  BIL T [D0] Below (N=102,104,102,100,101,102) | 0 | 0 | 0 | 0 | 0 | 0
  BIL T [D0] Within (N=102,104,102,100,101,102) | 101 | 102 | 100 | 98 | 99 | 101
  BIL T [D0] Above (N=102,104,102,100,101,102) | 1 | 2 | 1 | 1 | 1 | 1
  BIL T [D7] Below (N=102,101,100,99,100,99) | 0 | 0 | 0 | 0 | 0 | 0
  BIL T [D7] Within (N=102,101,100,99,100,99) | 101 | 100 | 97 | 98 | 99 | 97
  BIL T [D7] Above (N=102,101,100,99,100,99) | 1 | 1 | 3 | 1 | 1 | 2
  BIL T [D21] Below (N=101,100,97,97,99,99) | 0 | 0 | 0 | 0 | 0 | 0
  BIL T [D21] Within (N=101,100,97,97,99,99) | 99 | 97 | 95 | 96 | 97 | 97
  BIL T [D21] Above (N=101,100,97,97,99,99) | 2 | 3 | 2 | 1 | 2 | 1
  BIL T [D28] Below (N=101,98,96,98,98,97) | 0 | 0 | 0 | 0 | 0 | 0
  BIL T [D28] Within (N=101,98,96,98,98,97) | 99 | 96 | 94 | 95 | 97 | 95
  BIL T [D28] Above (N=101,98,96,98,98,97) | 1 | 2 | 2 | 2 | 1 | 1
  BIL T [D42] Below (N=101,97,95,95,96,97) | 0 | 0 | 0 | 0 | 0 | 0
  BIL T [D42] Within (N=101,97,95,95,96,97) | 98 | 93 | 92 | 91 | 93 | 95
  BIL T [D42] Above (N=101,97,95,95,96,97) | 3 | 4 | 2 | 4 | 1 | 2
  BIL T [D63] Below (N=100,95,95,95,97,97) | 0 | 0 | 0 | 0 | 0 | 0
  BIL T [D63] Within (N=100,95,95,95,97,97) | 98 | 92 | 92 | 94 | 93 | 94
  BIL T [D63] Above (N=100,95,95,95,97,97) | 1 | 2 | 2 | 1 | 3 | 1
  BIL T [D182] Below (N=99,91,88,91,93,97) | 0 | 0 | 0 | 0 | 0 | 0
  BIL T [D182] Within (N=99,91,88,91,93,97) | 99 | 87 | 86 | 89 | 90 | 96
  BIL T [D182] Above (N=99,91,88,91,93,97) | 0 | 3 | 2 | 2 | 2 | 1
  ALAT [D0] Unknown (N=102,101,102,100,101,102) | 0 | 0 | 1 | 1 | 1 | 0
  ALAT [D7] Unknown (N=102,101,100,99,100,99) | 0 | 0 | 0 | 0 | 0 | 0
  ALAT [D21] Unknown (N=101,100,97,97,99,99) | 0 | 0 | 0 | 0 | 0 | 1
  ALAT [D28] Unknown (N=101,98,96,98,98,97) | 1 | 0 | 0 | 1 | 0 | 1
  ALAT [D42] Unknown (N=101,97,95,95,96,97) | 0 | 0 | 1 | 0 | 2 | 0
  ALAT [D63] Unknown (N=100,95,95,95,97,97) | 1 | 1 | 1 | 0 | 1 | 2
  ALAT [D182] Unknown (N=99,91,88,91,93,97) | 0 | 1 | 0 | 0 | 1 | 0
  AP [D0] Unknown (N=102,104, 102,100,101,102) | 0 | 0 | 1 | 1 | 1 | 0
  AP [D7] Unknown (N=102,101,100,99,100,99) | 0 | 0 | 0 | 0 | 0 | 0
  AP [D21] Unknown (N=101,100,97,97,99,99) | 0 | 0 | 0 | 0 | 0 | 1
  AP [D28] Unknown (N=101,98,96,98,98,97) | 1 | 0 | 0 | 1 | 0 | 1
  AP [D42] Unknown (N=101,97, 95,95,96,97) | 0 | 0 | 1 | 0 | 2 | 0
  AP [D63] Unknown (N=100,95,95,95,97,97) | 1 | 1 | 1 | 0 | 1 | 2
  AP [D182] Unknown (N=99,91,88,91,93,97) | 0 | 1 | 0 | 0 | 1 | 0
  ASAT [D0] Unknown (N=102,104,102,100,101,102) | 0 | 0 | 1 | 1 | 1 | 0
  ASAT [D7] Unknown (N=102,101,100,99,100,99) | 0 | 0 | 1 | 0 | 0 | 0
  ASAT [D21] Unknown (N=101,100,97,97,99,99) | 0 | 0 | 0 | 0 | 0 | 1
  ASAT [D28] Unknown (N=101,98,96,98,98,97) | 1 | 0 | 0 | 1 | 0 | 1
  ASAT [D42] Unknown (N=101,97,95,95,96,97) | 0 | 0 | 1 | 0 | 2 | 0
  ASAT [D63] Unknown (N=100,95,95,95,97,97) | 1 | 1 | 2 | 0 | 2 | 2
  ASAT [D182] Unknown (N=99,91,88,91,93,97) | 1 | 1 | 1 | 0 | 1 | 0
  BAS [D0] Unknown (N=102,104,102,100,101,102) | 2 | 0 | 0 | 2 | 0 | 0
  BAS [D7] Unknown (N=102,101,100,99,100,99) | 0 | 1 | 0 | 1 | 0 | 0
  BAS [D21] Unknown (N=101,100,97,97,99,99) | 0 | 1 | 3 | 1 | 2 | 4
  BAS [D28] Unknown (N=101,98,96,98,98,97) | 2 | 2 | 0 | 2 | 1 | 3
  BAS [D42] Unknown (N=101,97,95,95,96,97) | 0 | 0 | 0 | 0 | 0 | 0
  BAS [D63] Unknown (N=100,95,95,95,97,97) | 0 | 0 | 0 | 0 | 0 | 0
  BAS [D182] Unknown (N=99,91,88,91,93,97) | 0 | 0 | 0 | 2 | 0 | 1
  BIL T [D0] Unknown (N=102,104,102,100,101,102) | 0 | 0 | 1 | 1 | 1 | 0
  BIL T [D7] Unknown (N=102,101,100,99,100,99) | 0 | 0 | 0 | 0 | 0 | 0
  BIL T [D21] Unknown (N=101,100,97,97,99,99) | 0 | 0 | 0 | 0 | 0 | 1
  BIL T [D28] Unknown (N=101,98,96,98,98,97) | 1 | 0 | 0 | 1 | 0 | 1
  BIL T [D42] Unknown (N=101,97,95,95,96,97) | 0 | 0 | 1 | 0 | 2 | 0
  BIL T [D63] Unknown (N=100,95,95,95,97,97) | 1 | 1 | 1 | 0 | 1 | 2
  BIL T [D182] Unknown (N=99,91,88,91,93,97) | 0 | 1 | 0 | 0 | 1 | 0

6. Secondary Outcome: Number of Subjects Reporting Clinical Laboratory Abnormalities in Biochemical and Haematological Parameters Assessed
Description: Laboratory parameters assessed were creatinine (CREA), bilirubin (BIL) (direct (D)), eosinophils (EOS), hemoglobin (Hgb), hematocrit (Hct). For each parameter and for each range it was assessed whether the values of the subjects were unknown, in above, below or within the range.
Time Frame: On Days 0, 7, 21, 28, 42, 63 and 182
Population: The Total Vaccinated cohort included all vaccinated subjects
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Number analyzed (Participants) | 102 | 104 | 102 | 100 | 101 | 102
Subjects
  BIL D [D0] Below (N=102,104,102,100,101,102) | 0 | 0 | 0 | 0 | 0 | 0
  BIL D [D0] Within (N=102,104,102,100,101,102) | 101 | 104 | 101 | 99 | 100 | 102
  BIL D [D0] Above (N=102,104,102,100,101,102) | 0 | 0 | 0 | 0 | 0 | 0
  BIL D [D0] Unknown (N=102,104,102,100,101,102) | 1 | 0 | 1 | 1 | 1 | 0
  BIL D [D7] Below (N=102,101,100,99,100,99) | 0 | 0 | 0 | 0 | 0 | 0
  BIL D [D7] Within (N=102,101,100,99,100,99) | 102 | 101 | 100 | 99 | 100 | 99
  BIL D [D7] Above (N=102,101,100,99,100,99) | 0 | 0 | 0 | 0 | 0 | 0
  BIL D [D7] Unknown(N=102,101,100,99,100,99) | 0 | 0 | 0 | 0 | 0 | 0
  BIL D [D21] Below (N=101,100,97,97,99,99) | 0 | 0 | 0 | 0 | 0 | 0
  BIL D [D21] Within (N=101,100,97,97,99,99) | 101 | 100 | 97 | 97 | 99 | 98
  BIL D [D21] Above (N=101,100,97,97,99,99) | 0 | 0 | 0 | 0 | 0 | 0
  BIL D [D21] Unknown (N=101,100,97,97,99,99) | 0 | 0 | 0 | 0 | 0 | 1
  BIL D [D28] Below (N=101,98,96,98,98,97) | 0 | 0 | 0 | 0 | 0 | 0
  BIL D [D28] Within (N=101,98,96,98,98,97) | 100 | 98 | 96 | 97 | 98 | 96
  BIL D [D28] Above (N=101,98,96,98,98,97) | 0 | 0 | 0 | 0 | 0 | 0
  BIL D [D28] Unknown (N=101,98,96,98,98,97) | 1 | 0 | 0 | 1 | 0 | 1
  BIL D [D42] Below (N=101,97,95,95,96,97) | 0 | 0 | 0 | 0 | 0 | 0
  BIL D [D42] Within (N=101,97,95,95,96,97) | 101 | 97 | 94 | 95 | 94 | 97
  BIL D [D42] Above (N=101,97,95,95,96,97) | 0 | 0 | 0 | 0 | 0 | 0
  BIL D [D42] Unknown (N=101,97,95,95,96,97) | 0 | 0 | 1 | 0 | 2 | 0
  BIL D [D63] Below (N=100,95,95,95,97,97) | 0 | 0 | 0 | 0 | 0 | 0
  BIL D [D63] Within (N=100,95,95,95,97,97) | 99 | 94 | 94 | 95 | 96 | 95
  BIL D [D63] Above (N=100,95,95,95,97,97) | 0 | 0 | 0 | 0 | 0 | 0
  BIL D [D63] Unknown (N=100,95,95,95,97,97) | 1 | 1 | 1 | 0 | 1 | 2
  BIL D [D182] Below (N=99,91,88,91,93,97) | 0 | 0 | 0 | 0 | 0 | 0
  BIL D [D182] Within (N=99,91,88,91,93,97) | 99 | 90 | 88 | 91 | 92 | 96
  BIL D [D182] Above (N=99,91,88,91,93,97) | 0 | 0 | 0 | 0 | 0 | 1
  BIL D [D182] Unknown (N=99,91,88,91,93,97) | 0 | 1 | 0 | 0 | 1 | 0
  CREA [D0] Below (N=102,104,102,100,101,102) | 8 | 6 | 6 | 9 | 8 | 9
  CREA [D0] Within (N=102,104,102,100,101,102) | 93 | 97 | 94 | 88 | 92 | 92
  CREA [D0] Above (N=102,104,102,100,101,102) | 1 | 1 | 1 | 2 | 0 | 1
  CREA [D0] Unknown (N=102,104,102,100,101,102) | 0 | 0 | 1 | 1 | 1 | 0
  CREA [D7] Below (N=102,101,100,99,100,99) | 8 | 6 | 9 | 17 | 7 | 8
  CREA [D7] Within (N=102,101,100,99,100,99) | 94 | 93 | 91 | 81 | 93 | 90
  CREA [D7] Above (N=102,101,100,99,100,99) | 0 | 2 | 0 | 1 | 0 | 1
  CREA [D7] Unknown (N=102,101,100,99,100,99) | 0 | 0 | 0 | 0 | 0 | 0
  CREA [D21] Below (N=101,100,97,97,99,99) | 12 | 6 | 5 | 16 | 10 | 9
  CREA [D21] Within (N=101,100,97,97,99,99) | 88 | 92 | 92 | 81 | 89 | 87
  CREA [D21] Above (N=101,100,97,97,99,99) | 1 | 2 | 0 | 0 | 0 | 2
  CREA [D21] Unknown (N=101,100,97,97,99,99) | 0 | 0 | 0 | 0 | 0 | 1
  CREA [D28] Below (N=101,98,96,98,98,97) | 5 | 8 | 6 | 15 | 7 | 7
  CREA [D28] Within (N=101,98,96,98,98,97) | 95 | 90 | 89 | 81 | 91 | 89
  CREA [D28] Above (N=101,98,96,98,98,97) | 0 | 0 | 1 | 1 | 0 | 0
  CREA [D28] Unknown (N=101,98,96,98,98,97) | 1 | 0 | 0 | 1 | 0 | 1
  CREA [D42] Below (N=101,97,95,95,96,97) | 6 | 5 | 5 | 10 | 9 | 11
  CREA [D42] Within (N=101,97,95,95,96,97) | 95 | 90 | 88 | 84 | 85 | 86
  CREA [D42] Above (N=101,97,95,95,96,97) | 0 | 2 | 1 | 1 | 0 | 0
  CREA [D42] Unknown (N=101,97,95,95,96,97) | 0 | 0 | 1 | 0 | 2 | 0
  CREA [D63] Below (N=100,95,95,95,97,97) | 7 | 7 | 7 | 14 | 7 | 9
  CREA [D63] Within (N=100,95,95,95,97,97) | 92 | 86 | 87 | 78 | 89 | 85
  CREA [D63] Above (N=100,95,95,95,97,97) | 0 | 1 | 0 | 3 | 0 | 1
  CREA [D63] Unknown (N=100,95,95,95,97,97) | 1 | 1 | 1 | 0 | 1 | 2
  CREA [D182] Below (N=99,91,88,91,93,97) | 14 | 7 | 7 | 10 | 6 | 14
  CREA [D182] Within (N=99,91,88,91,93,97) | 84 | 82 | 80 | 81 | 86 | 83
  CREA [D182] Above (N=99,91,88,91,93,97) | 1 | 1 | 1 | 0 | 0 | 0
  CREA [D182] Unknown (N=99,91,88,91,93,97) | 0 | 1 | 0 | 0 | 1 | 0
  EOS [D0] Below (N=102,104,102,100,101,102) | 2 | 6 | 7 | 5 | 9 | 5
  EOS [D0] Within (N=102,104,102,100,101,102) | 97 | 96 | 93 | 92 | 90 | 97
  EOS [D0] Above (N=102,104,102,100,101,102) | 1 | 2 | 2 | 1 | 2 | 0
  EOS [D0] Unknown (N=102,104,102,100,101,102) | 2 | 0 | 0 | 2 | 0 | 0
  EOS [D7] Below (N=102,101,100,99,100,99) | 7 | 4 | 7 | 1 | 5 | 8
  EOS [D7] Within (N=102,101,100,99,100,99) | 93 | 93 | 91 | 95 | 92 | 89
  EOS [D7] Above (N=102,101,100,99,100,99) | 2 | 3 | 2 | 2 | 3 | 2
  EOS [D7] Unknown (N=102,101,100,99,100,99) | 0 | 1 | 0 | 1 | 0 | 0
  EOS [D21] Below (N=101,100,97,97,99,99) | 2 | 8 | 9 | 8 | 9 | 3
  EOS [D21] Within (N=101,100,97,97,99,99) | 97 | 87 | 85 | 87 | 85 | 92
  EOS [D21] Above (N=101,100,97,97,99,99) | 2 | 4 | 0 | 1 | 3 | 0
  EOS [D21] Unknown (N=101,100,97,97,99,99) | 0 | 1 | 3 | 1 | 2 | 4
  EOS [D28] Below (N=101,98,96,98,98,97) | 4 | 4 | 7 | 2 | 7 | 5
  EOS [D28] Within (N=101,98,96,98,98,97) | 94 | 90 | 89 | 93 | 90 | 87
  EOS [D28] Above (N=101,98,96,98,98,97) | 1 | 2 | 0 | 1 | 0 | 2
  EOS [D28] Unknown (N=101,98,96,98,98,97) | 2 | 2 | 0 | 2 | 1 | 3
  EOS [D42] Below (N=101,97,95,95,96,97) | 4 | 9 | 6 | 5 | 8 | 9
  EOS [D42] Within (N=101,97,95,95,96,97) | 96 | 86 | 89 | 89 | 85 | 88
  EOS [D42] Above (N=101,97,95,95,96,97) | 1 | 2 | 0 | 1 | 3 | 0
  EOS [D42] Unknown (N=101,97,95,95,96,97) | 0 | 0 | 0 | 0 | 0 | 0
  EOS [D63] Below (N=100,95,95,95,97,97) | 2 | 9 | 8 | 4 | 8 | 10
  EOS [D63] Within (N=100,95,95,95,97,97) | 97 | 82 | 85 | 90 | 88 | 86
  EOS [D63] Above (N=100,95,95,95,97,97) | 1 | 4 | 2 | 1 | 1 | 1
  EOS [D63] Unknown (N=100,95,95,95,97,97) | 0 | 0 | 0 | 0 | 0 | 0
  EOS [D182] Below (N=99,91,88,91,93,97) | 3 | 4 | 9 | 3 | 6 | 5
  EOS [D182] Within (N=99,91,88,91,93,97) | 94 | 86 | 78 | 83 | 84 | 89
  EOS [D182] Above (N=99,91,88,91,93,97) | 2 | 1 | 1 | 3 | 3 | 2
  EOS [D182] Unknown (N=99,91,88,91,93,97) | 0 | 0 | 0 | 2 | 0 | 1
  Hct [D0] Below (N=102,104,102,100,101,102) | 4 | 2 | 4 | 3 | 3 | 5
  Hct [D0] Within (N=102,104,102,100,101,102) | 94 | 99 | 95 | 92 | 97 | 97
  Hct [D0] Above (N=102,104,102,100,101,102) | 2 | 3 | 3 | 3 | 1 | 0
  Hct [D0] Unknown (N=102,104,102,100,101,102) | 2 | 0 | 0 | 2 | 0 | 0
  Hct [D7] Below (N=102,101,100,99,100,99) | 7 | 7 | 4 | 4 | 3 | 6
  Hct [D7] Within (N=102,101,100,99,100,99) | 93 | 91 | 95 | 92 | 97 | 92
  Hct [D7] Above (N=102,101,100,99,100,99) | 2 | 2 | 1 | 2 | 0 | 1
  Hct [D7] Unknown (N=102,101,100,99,100,99) | 0 | 1 | 0 | 1 | 0 | 0
  Hct [D21] Below (N=101,100,97,97,99,99) | 8 | 4 | 5 | 8 | 6 | 4
  Hct [D21] Within (N=101,100,97,97,99,99) | 92 | 94 | 88 | 88 | 91 | 91
  Hct [D21] Above (N=101,100,97,97,99,99) | 1 | 1 | 1 | 0 | 0 | 1
  Hct [D21] Unknown (N=101,100,97,97,99,99) | 0 | 1 | 3 | 1 | 2 | 3
  Hct [D28] Below (N=101,98,96,98,98,97) | 10 | 6 | 8 | 9 | 5 | 9
  Hct [D28] Within (N=101,98,96,98,98,97) | 89 | 88 | 86 | 88 | 92 | 84
  Hct [D28] Above (N=101,98,96,98,98,97) | 1 | 2 | 2 | 0 | 0 | 1
  Hct [D28] Unknown (N=101,98,96,98,98,97) | 1 | 2 | 0 | 1 | 1 | 3
  Hct [D42] Below (N=101,97,95,95,96,97) | 11 | 9 | 9 | 7 | 10 | 14
  Hct [D42] Within (N=101,97,95,95,96,97) | 90 | 86 | 86 | 88 | 86 | 83
  Hct [D42] Above (N=101,97,95,95,96,97) | 0 | 2 | 0 | 0 | 0 | 0
  Hct [D42] Unknown (N=101,97,95,95,96,97) | 0 | 0 | 0 | 0 | 0 | 0
  Hct [D63] Below (N=100,95,95,95,97,97) | 8 | 10 | 11 | 6 | 10 | 10
  Hct [D63] Within (N=100,95,95,95,97,97) | 92 | 84 | 84 | 89 | 87 | 87
  Hct [D63] Above (N=100,95,95,95,97,97) | 0 | 1 | 0 | 0 | 0 | 0
  Hct [D63] Unknown (N=100,95,95,95,97,97) | 0 | 0 | 0 | 0 | 0 | 0
  Hct [D182] Below (N=99,91,88,91,93,97) | 4 | 6 | 4 | 3 | 7 | 10
  Hct [D182] Within (N=99,91,88,91,93,97) | 93 | 84 | 82 | 85 | 86 | 86
  Hct [D182] Above (N=99,91,88,91,93,97) | 2 | 1 | 2 | 1 | 0 | 1
  Hct [D182] Unknown (N=99,91,88,91,93,97) | 0 | 0 | 0 | 2 | 0 | 0
  Hgb [D0] Below (N=102,104,102,100,101,102) | 2 | 6 | 5 | 1 | 4 | 5
  Hgb [D0] Within (N=102,104,102,100,101,102) | 97 | 97 | 95 | 97 | 97 | 97
  Hgb [D0] Above (N=102,104,102,100,101,102) | 1 | 1 | 2 | 0 | 0 | 0
  Hgb [D0] Unknown (N=102,104,102,100,101,102) | 2 | 0 | 0 | 2 | 0 | 0
  Hgb [D7] Below (N=102,101,100,99,100,99) | 6 | 7 | 5 | 2 | 4 | 3
  Hgb [D7] Within (N=102,101,100,99,100,99) | 94 | 91 | 94 | 96 | 96 | 95
  Hgb [D7] Above (N=102,101,100,99,100,99) | 2 | 2 | 1 | 0 | 0 | 1
  Hgb [D7] Unknown (N=102,101,100,99,100,99) | 0 | 1 | 0 | 1 | 0 | 0
  Hgb [D21] Below (N=101,100,97,97,99,99) | 6 | 5 | 3 | 6 | 5 | 4
  Hgb [D21] Within (N=101,100,97,97,99,99) | 93 | 94 | 90 | 90 | 92 | 91
  Hgb [D21] Above (N=101,100,97,97,99,99) | 2 | 0 | 1 | 0 | 0 | 1
  Hgb [D21] Unknown (N=101,100,97,97,99,99) | 0 | 1 | 3 | 1 | 2 | 3
  Hgb [D28] Below (N=101,98,96,98,98,97) | 10 | 7 | 5 | 8 | 1 | 4
  Hgb [D28] Within (N=101,98,96,98,98,97) | 90 | 88 | 89 | 89 | 96 | 90
  Hgb [D28] Above (N=101,98,96,98,98,97) | 0 | 1 | 2 | 0 | 0 | 0
  Hgb [D28] Unknown (N=101,98,96,98,98,97) | 1 | 2 | 0 | 1 | 1 | 3
  Hgb [D42] Below (N=101,97,95,95,96,97) | 7 | 8 | 6 | 3 | 6 | 11
  Hgb [D42] Within (N=101,97,95,95,96,97) | 94 | 87 | 89 | 92 | 90 | 86
  Hgb [D42] Above (N=101,97,95,95,96,97) | 0 | 2 | 0 | 0 | 0 | 0
  Hgb [D42] Unknown (N=101,97,95,95,96,97) | 0 | 0 | 0 | 0 | 0 | 0
  Hgb [D63] Below (N=100,95,95,95,97,97) | 8 | 10 | 6 | 4 | 9 | 10
  Hgb [D63] Within (N=100,95,95,95,97,97) | 92 | 83 | 89 | 91 | 88 | 87
  Hgb [D63] Above (N=100,95,95,95,97,97) | 0 | 2 | 0 | 0 | 0 | 0
  Hgb [D63] Unknown (N=100,95,95,95,97,97) | 0 | 0 | 0 | 0 | 0 | 0
  Hgb [D182] Below (N=99,91,88,91,93,97) | 9 | 6 | 5 | 5 | 6 | 9
  Hgb [D182] Within (N=99,91,88,91,93,97) | 89 | 84 | 81 | 84 | 87 | 87
  Hgb [D182] Above (N=99,91,88,91,93,97) | 1 | 1 | 2 | 0 | 0 | 1
  Hgb [D182] Unknown (N=99,91,88,91,93,97) | 0 | 0 | 0 | 2 | 0 | 0

7. Secondary Outcome: Number of Subjects Reporting Solicited Local Symptoms.
Description: Solicited local symptoms assessed were pain, redness and swelling
Time Frame: During a 7-day follow-up period (Days 0-6) post-vaccination period
Population: The Total Vaccinated cohort included all vaccinated subjects
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Number analyzed (Participants) | 102 | 100 | 100 | 99 | 101 | 100
Subjects
  Pain | 75 | 89 | 66 | 94 | 69 | 95
  Redness | 2 | 6 | 1 | 5 | 1 | 11
  Swelling | 2 | 15 | 2 | 9 | 0 | 16

8. Secondary Outcome: Number of Subjects Reporting Solicited General Symptoms.
Description: Solicited general symptoms assessed were fatigue, headache, joint pain at other location, muscle aches, shivering, sweating and temperature. Temperature is defined as an axillary temperature equal to or above 38.0 degrees Celsius (°C).
Time Frame: During a 7-day follow-up period (Days 0-6) post-vaccination period
Population: The Total Vaccinated cohort included all vaccinated subjects
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Number analyzed (Participants) | 102 | 100 | 100 | 99 | 101 | 100
Subjects
  Fatigue | 54 | 62 | 41 | 58 | 57 | 56
  Headache | 52 | 58 | 51 | 51 | 49 | 54
  Joint pain at other location | 24 | 34 | 24 | 28 | 26 | 23
  Muscle aches | 38 | 52 | 39 | 53 | 43 | 54
  Shivering | 21 | 30 | 19 | 24 | 21 | 25
  Sweating | 22 | 21 | 21 | 17 | 12 | 25
  Temperature (axillary) >=38°C | 3 | 9 | 3 | 2 | 1 | 4

9. Secondary Outcome: Number of Subjects Reporting Clinical Laboratory Abnormalities in Biochemical and Haematological Parameters Assessed
Description: Laboratory parameters assessed were serum urea nitrogen (SUN), white blood cells (WBC), red blood cells (RBC). For each parameter and for each range it was assessed whether the values of the subjects were unknown, above, below or within the range.
Time Frame: On Days 0, 7, 21, 28, 42, 63 and 182
Population: The Total Vaccinated cohort included all vaccinated subjects
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Number analyzed (Participants) | 102 | 104 | 102 | 100 | 101 | 102
Subjects
  RBC [D0] Below (N=102,104,102,100101,102) | 4 | 2 | 7 | 3 | 2 | 4
  RBC [D0] Within (N=102,104,102,100101,102) | 96 | 100 | 95 | 93 | 99 | 98
  RBC [D0] Above (N=102,104,102,100101,102) | 0 | 2 | 0 | 2 | 0 | 0
  RBC [D0] Unknown (N=102,104,102,100101,102) | 2 | 0 | 0 | 2 | 0 | 0
  RBC [D7] Below (N=102,101,100,99,100,99) | 3 | 5 | 5 | 4 | 5 | 3
  RBC [D7] Within (N=102,101,100,99,100,99) | 99 | 94 | 95 | 93 | 95 | 96
  RBC [D7] Above (N=102,101,100,99,100,99) | 0 | 1 | 0 | 1 | 0 | 0
  RBC [D7] Unknown (N=102,101,100,99,100,99) | 0 | 1 | 0 | 1 | 0 | 0
  RBC [D21] Below (N=101,100,97,97,99,99) | 5 | 7 | 5 | 6 | 3 | 6
  RBC [D21] Within (N=101,100,97,97,99,99) | 96 | 92 | 89 | 90 | 94 | 90
  RBC [D21] Above (N=101,100,97,97,99,99) | 0 | 0 | 0 | 0 | 0 | 0
  RBC [D21] Unknown (N=101,100,97,97,99,99) | 0 | 1 | 3 | 1 | 2 | 3
  RBC [D28] Below (N=101,98,96,98,98,97) | 5 | 8 | 8 | 7 | 2 | 8
  RBC [D28] Within (N=101,98,96,98,98,97) | 95 | 87 | 88 | 89 | 95 | 86
  RBC [D28] Above (N=101,98,96,98,98,97) | 0 | 1 | 0 | 1 | 0 | 0
  RBC [D28] Unknown (N=101,98,96,98,98,97) | 1 | 2 | 0 | 1 | 1 | 3
  RBC [D42] Below (N=101,97,95,95,96,97) | 2 | 9 | 9 | 6 | 7 | 12
  RBC [D42] Within (N=101,97,95,95,96,97) | 99 | 87 | 86 | 89 | 89 | 85
  RBC [D42] Above (N=101,97,95,95,96,97) | 0 | 1 | 0 | 0 | 0 | 0
  RBC [D42] Unknown (N=101,97,95,95,96,97) | 0 | 0 | 0 | 0 | 0 | 0
  RBC [D63] Below (N=100,95,95,95,97,97) | 6 | 8 | 5 | 5 | 6 | 12
  RBC [D63] Within (N=100,95,95,95,97,97) | 94 | 86 | 90 | 89 | 91 | 85
  RBC [D63] Above (N=100,95,95,95,97,97) | 0 | 1 | 0 | 1 | 0 | 0
  RBC [D63] Unknown (N=100,95,95,95,97,97) | 0 | 0 | 0 | 0 | 0 | 0
  RBC [D182] Below (N=99,91,88,91,93,97) | 6 | 6 | 9 | 4 | 5 | 10
  RBC [D182] Within (N=99,91,88,91,93,97) | 92 | 85 | 77 | 84 | 88 | 87
  RBC [D182] Above (N=99,91,88,91,93,97) | 1 | 0 | 2 | 1 | 0 | 0
  RBC [D182] Unknown (N=99,91,88,91,93,97) | 0 | 0 | 0 | 2 | 0 | 0
  SUN [D0] Below (N=102,104,102,100101,102) | 1 | 0 | 1 | 1 | 1 | 2
  SUN [D0] Within (N=102,104,102,100101,102) | 100 | 104 | 100 | 98 | 98 | 99
  SUN [D0] Above (N=102,104,102,100101,102) | 1 | 0 | 0 | 0 | 1 | 1
  SUN [D0] Unknown (N=102,104,102,100101,102) | 0 | 0 | 1 | 1 | 1 | 0
  SUN [D7] Below (N=102,101,100,99,100,99) | 2 | 1 | 4 | 1 | 0 | 0
  SUN [D7] Within (N=102,101,100,99,100,99) | 100 | 99 | 96 | 98 | 99 | 99
  SUN [D7] Above (N=102,101,100,99,100,99) | 0 | 1 | 0 | 0 | 1 | 0
  SUN [D7] Unknown (N=102,101,100,99,100,99) | 0 | 0 | 0 | 0 | 0 | 0
  SUN [D21] Below (N=101,100,97,97,99,99) | 1 | 1 | 0 | 2 | 1 | 3
  SUN [D21] Within (N=101,100,97,97,99,99) | 100 | 99 | 96 | 95 | 98 | 95
  SUN [D21] Above (N=101,100,97,97,99,99) | 0 | 0 | 1 | 0 | 0 | 0
  SUN [D21] Unknown (N=101,100,97,97,99,99) | 0 | 0 | 0 | 0 | 0 | 1
  SUN [D28] Below (N=101,98,96,98,98,97) | 2 | 1 | 0 | 0 | 0 | 4
  SUN [D28] Within (N=101,98,96,98,98,97) | 98 | 97 | 96 | 97 | 98 | 91
  SUN [D28] Above (N=101,98,96,98,98,97) | 0 | 0 | 0 | 0 | 0 | 1
  SUN [D28] Unknown (N=101,98,96,98,98,97) | 1 | 0 | 0 | 1 | 0 | 1
  SUN [D42] Below (N=101,97,95,95,96,97) | 1 | 1 | 2 | 1 | 2 | 2
  SUN [D42] Within (N=101,97,95,95,96,97) | 100 | 96 | 91 | 94 | 92 | 95
  SUN [D42] Above (N=101,97,95,95,96,97) | 0 | 0 | 1 | 0 | 0 | 0
  SUN [D42] Unknown (N=101,97,95,95,96,97) | 0 | 0 | 1 | 0 | 2 | 0
  SUN [D63] Below (N=100,95,95,95,97,97) | 1 | 0 | 1 | 2 | 0 | 1
  SUN [D63] Within (N=100,95,95,95,97,97) | 98 | 94 | 93 | 93 | 96 | 94
  SUN [D63] Above (N=100,95,95,95,97,97) | 0 | 0 | 0 | 0 | 0 | 0
  SUN [D63] Unknown (N=100,95,95,95,97,97) | 1 | 1 | 1 | 0 | 1 | 2
  SUN [D182] Below (N=99,91,88,91,93,97) | 0 | 2 | 1 | 1 | 1 | 3
  SUN [D182] Within (N=99,91,88,91,93,97) | 99 | 88 | 87 | 90 | 91 | 94
  SUN [D182] Above (N=99,91,88,91,93,97) | 0 | 0 | 0 | 0 | 0 | 0
  SUN [D182] Unknown (N=99,91,88,91,93,97) | 0 | 1 | 0 | 0 | 1 | 0
  WBC [D0] Below (N=102,104,102,100,101,102) | 1 | 2 | 5 | 3 | 2 | 2
  WBC [D0] Within (N=102,104,102,100,101,102) | 95 | 100 | 94 | 93 | 95 | 95
  WBC [D0] Above (N=102,104,102,100,101,102) | 4 | 2 | 3 | 2 | 4 | 5
  WBC [D0] Unknown (N=102,104,102,100,101,102) | 2 | 0 | 0 | 2 | 0 | 0
  WBC [D7] Below (N=102,101,100,99,100,99) | 3 | 0 | 2 | 1 | 3 | 2
  WBC [D7] Within (N=102,101,100,99,100,99) | 99 | 97 | 98 | 92 | 94 | 94
  WBC [D7] Above (N=102,101,100,99,100,99) | 0 | 3 | 0 | 5 | 3 | 3
  WBC [D7] Unknown (N=102,101,100,99,100,99) | 0 | 1 | 0 | 1 | 0 | 0
  WBC [D21] Below (N=101,100,97,97,99,99) | 1 | 4 | 2 | 2 | 3 | 2
  WBC [D21] Within (N=101,100,97,97,99,99) | 98 | 94 | 90 | 93 | 91 | 90
  WBC [D21] Above (N=101,100,97,97,99,99) | 2 | 1 | 2 | 1 | 3 | 3
  WBC [D21] Unknown (N=101,100,97,97,99,99) | 0 | 1 | 3 | 1 | 2 | 4
  WBC [D28] Below (N=101,98,96,98,98,97) | 0 | 1 | 3 | 3 | 2 | 0
  WBC [D28] Within (N=101,98,96,98,98,97) | 98 | 92 | 92 | 92 | 93 | 91
  WBC [D28] Above (N=101,98,96,98,98,97) | 1 | 3 | 1 | 1 | 2 | 3
  WBC [D28] Unknown (N=101,98,96,98,98,97) | 2 | 2 | 0 | 2 | 1 | 3
  WBC [D42] Below (N=101,97,95,95,96,97) | 0 | 4 | 2 | 3 | 3 | 3
  WBC [D42] Within (N=101,97,95,95,96,97) | 100 | 91 | 92 | 90 | 92 | 91
  WBC [D42] Above (N=101,97,95,95,96,97) | 1 | 2 | 1 | 2 | 1 | 3
  WBC [D42] Unknown (N=101,97,95,95,96,97) | 0 | 0 | 0 | 0 | 0 | 0
  WBC [D63] Below (N=100,95,95,95,97,97) | 1 | 2 | 1 | 2 | 3 | 3
  WBC [D63] Within (N=100,95,95,95,97,97) | 98 | 92 | 93 | 89 | 91 | 91
  WBC [D63] Above (N=100,95,95,95,97,97) | 1 | 1 | 1 | 4 | 3 | 3
  WBC [D63] Unknown (N=100,95,95,95,97,97) | 0 | 0 | 0 | 0 | 0 | 0
  WBC [D182] Below (N=99,91,88,91,93,97) | 2 | 2 | 4 | 3 | 2 | 4
  WBC [D182] Within (N=99,91,88,91,93,97) | 93 | 87 | 82 | 84 | 88 | 91
  WBC [D182] Above (N=99,91,88,91,93,97) | 4 | 2 | 2 | 2 | 3 | 1
  WBC [D182] Unknown (N=99,91,88,91,93,97) | 0 | 0 | 0 | 2 | 0 | 1

10. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs).
Description: An unsolicited adverse event is any adverse event (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: Within the 84-day (Days 0-83) post-vaccination period.
Population: The Total Vaccinated Cohort included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Number analyzed (Participants) | 102 | 104 | 102 | 100 | 101 | 102
Subjects | 68 | 65 | 57 | 57 | 62 | 63

11. Secondary Outcome: Number of Subjects Reporting Medically Attended Visits (MAEs).
Description: The day 368 was the last contact day for the last subject reporting the event. For each solicited and unsolicited symptom the subject experienced, the subject was asked if they received medical attention defined as hospitalization, an emergency room visit or a visit to or from medical personnel for any reason.
Time Frame: During the entire study period (Days 0-368).
Population: The Total Vaccinated Cohort included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Number analyzed (Participants) | 102 | 104 | 102 | 100 | 101 | 102
Subjects | 51 | 42 | 40 | 42 | 38 | 45

12. Secondary Outcome: Number of Subjects Reporting Potential Immune Diseases (pIMDs).
Description: The day 406 was the last contact day with the subjects reporting the event. Potential immune-mediated diseases (pIMDs) are a subset of AEs that include both clearly autoimmune diseases and also other inflammatory and/or neurologic disorders which may or may not have an autoimmune etiology.
Time Frame: During the entire study period (Days 0-406).
Population: The Total Vaccinated Cohort included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Number analyzed (Participants) | 102 | 104 | 102 | 100 | 101 | 102
Subjects | 0 | 0 | 0 | 0 | 0 | 1

13. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs).
Description: The day 329 was the last contact day with the subjects reporting serious adverse events.
  SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subjects.
Time Frame: During the entire study period (Days 0-329).
Population: The Total Vaccinated Cohort included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Number analyzed (Participants) | 102 | 104 | 102 | 100 | 101 | 102
Subjects | 3 | 1 | 1 | 2 | 1 | 3

14. Secondary Outcome: Number of Subjects Reporting Clinical Laboratory Abnormalities in Biochemical and Haematological Parameters Assessed
Description: Laboratory parameters assessed were neutrophils (NEU), lymphocytes (LYM), monocytes (MON) and platelets (PLA). For each parameter and for each range it was assessed whether the values of the subjects were unknown, in above, below or within the range.
Time Frame: On Days 0, 7, 21, 28, 42, 63 and 182
Population: The Total Vaccinated cohort included all vaccinated subjects
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Number analyzed (Participants) | 102 | 104 | 102 | 100 | 101 | 102
Subjects
  LYM [D0] Below (N=102,104,102,100,101,102) | 0 | 2 | 0 | 0 | 0 | 0
  LYM [D0] Within (N=102,104,102,100,101,102) | 100 | 101 | 102 | 98 | 101 | 101
  LYM [D0] Above (N=102,104,102,100,101,102) | 0 | 1 | 0 | 0 | 0 | 1
  LYM [D0] Unknown (N=102,104,102,100,101,102) | 2 | 0 | 0 | 2 | 0 | 0
  LYM [D7] Below (N=102,101,100,99,100,99) | 1 | 0 | 1 | 0 | 0 | 1
  LYM [D7] Within (N=102,101,100,99,100,99) | 100 | 100 | 99 | 98 | 100 | 98
  LYM [D7] Above (N=102,101,100,99,100,99) | 1 | 0 | 0 | 0 | 0 | 0
  LYM [D7] Unknown (N=102,101,100,99,100,99) | 0 | 1 | 0 | 1 | 0 | 0
  LYM [D21] Below (N=101,100,97,97,99,99) | 0 | 1 | 0 | 0 | 0 | 0
  LYM [D21] Within (N=101,100,97,97,99,99) | 101 | 98 | 94 | 95 | 97 | 94
  LYM [D21] Above (N=101,100,97,97,99,99) | 0 | 0 | 0 | 1 | 0 | 1
  LYM [D21] Unknown (N=101,100,97,97,99,99) | 0 | 1 | 3 | 1 | 2 | 4
  LYM [D28] Below (N=101,98,96,98,98,97) | 0 | 0 | 0 | 0 | 0 | 0
  LYM [D28] Within (N=101,98,96,98,98,97) | 99 | 96 | 95 | 96 | 97 | 93
  LYM [D28] Above (N=101,98,96,98,98,97) | 0 | 0 | 1 | 0 | 0 | 1
  LYM [D28] Unknown (N=101,98,96,98,98,97) | 2 | 2 | 0 | 2 | 1 | 3
  LYM [D42] Below (N=101,97,95,95,96,97) | 0 | 2 | 0 | 0 | 3 | 0
  LYM [D42] Within (N=101,97,95,95,96,97) | 101 | 95 | 95 | 94 | 93 | 97
  LYM [D42] Above (N=101,97,95,95,96,97) | 0 | 0 | 0 | 1 | 0 | 0
  LYM [D42] Unknown (N=101,97,95,95,96,97) | 0 | 0 | 0 | 0 | 0 | 0
  LYM [D63] Below (N=100,95,95,95,97,97) | 0 | 0 | 0 | 0 | 1 | 0
  LYM [D63] Within (N=100,95,95,95,97,97) | 100 | 95 | 95 | 95 | 96 | 96
  LYM [D63] Above (N=100,95,95,95,97,97) | 0 | 0 | 0 | 0 | 0 | 1
  LYM [D63] Unknown (N=100,95,95,95,97,97) | 0 | 0 | 0 | 0 | 0 | 0
  LYM [D182] Below (N=99,91,88,91,93,97) | 0 | 1 | 0 | 0 | 1 | 0
  LYM [D182] Within (N=99,91,88,91,93,97) | 98 | 90 | 88 | 89 | 91 | 95
  LYM [D182] Above (N=99,91,88,91,93,97) | 1 | 0 | 0 | 0 | 1 | 1
  LYM [D182] Unknown (N=99,91,88,91,93,97) | 0 | 0 | 0 | 2 | 0 | 1
  MON [D0] Below (N=102,104,102,100,101,102) | 11 | 18 | 26 | 18 | 13 | 23
  MON [D0] Within (N=102,104,102,100,101,102) | 89 | 86 | 75 | 79 | 88 | 79
  MON [D0] Above (N=102,104,102,100,101,102) | 0 | 0 | 1 | 1 | 0 | 0
  MON [D0] Unknown (N=102,104,102,100,101,102) | 2 | 0 | 0 | 2 | 0 | 0
  MON [D7] Below (N=102,101,100,99,100,99) | 20 | 14 | 22 | 12 | 13 | 22
  MON [D7] Within (N=102,101,100,99,100,99) | 82 | 86 | 78 | 86 | 87 | 77
  MON [D7] Above (N=102,101,100,99,100,99) | 0 | 0 | 0 | 0 | 0 | 0
  MON [D7] Unknown (N=102,101,100,99,100,99) | 0 | 1 | 0 | 1 | 0 | 0
  MON [D21] Below (N=101,100,97,97,99,99) | 25 | 20 | 20 | 12 | 18 | 20
  MON [D21] Within (N=101,100,97,97,99,99) | 76 | 79 | 74 | 84 | 79 | 75
  MON [D21] Above (N=101,100,97,97,99,99) | 0 | 0 | 0 | 0 | 0 | 0
  MON [D21] Unknown (N=101,100,97,97,99,99) | 0 | 1 | 3 | 1 | 2 | 4
  MON [D28] Below (N=101,98,96,98,98,97) | 17 | 19 | 26 | 26 | 17 | 19
  MON [D28] Within (N=101,98,96,98,98,97) | 82 | 77 | 70 | 70 | 80 | 75
  MON [D28] Above (N=101,98,96,98,98,97) | 0 | 0 | 0 | 0 | 0 | 0
  MON [D28] Unknown (N=101,98,96,98,98,97) | 2 | 2 | 0 | 2 | 1 | 3
  MON [D42] Below (N=101,97,95,95,96,97) | 16 | 19 | 20 | 25 | 20 | 20
  MON [D42] Within (N=101,97,95,95,96,97) | 85 | 78 | 75 | 70 | 76 | 77
  MON [D42] Above (N=101,97,95,95,96,97) | 0 | 0 | 0 | 0 | 0 | 0
  MON [D42] Unknown (N=101,97,95,95,96,97) | 0 | 0 | 0 | 0 | 0 | 0
  MON [D63] Below (N=100,95,95,95,97,97) | 17 | 20 | 21 | 19 | 15 | 18
  MON [D63] Within (N=100,95,95,95,97,97) | 82 | 75 | 73 | 76 | 82 | 79
  MON [D63] Above (N=100,95,95,95,97,97) | 1 | 0 | 1 | 0 | 0 | 0
  MON [D63] Unknown (N=100,95,95,95,97,97) | 0 | 0 | 0 | 0 | 0 | 0
  MON [D182] Below (N=99,91,88,91,93,97) | 17 | 20 | 20 | 21 | 20 | 23
  MON [D182] Within (N=99,91,88,91,93,97) | 82 | 71 | 68 | 68 | 73 | 73
  MON [D182] Above (N=99,91,88,91,93,97) | 0 | 0 | 0 | 0 | 0 | 0
  MON [D182] Unknown (N=99,91,88,91,93,97) | 0 | 0 | 0 | 2 | 0 | 1
  NEU [D0] Below (N=102,104,102,100,101,102) | 1 | 4 | 4 | 4 | 0 | 4
  NEU [D0] Within (N=102,104,102,100,101,102) | 98 | 98 | 97 | 92 | 98 | 93
  NEU [D0] Above (N=102,104,102,100,101,102) | 1 | 2 | 1 | 2 | 3 | 5
  NEU [D0] Unknown (N=102,104,102,100,101,102) | 2 | 0 | 0 | 2 | 0 | 0
  NEU [D7] Below (N=101,100,98,97,97,97) | 2 | 2 | 2 | 2 | 1 | 3
  NEU [D7] Within (N=101,100,98,97,97,97) | 96 | 94 | 94 | 90 | 93 | 91
  NEU [D7] Above (N=101,100,98,97,97,97) | 3 | 3 | 2 | 4 | 3 | 3
  NEU [D7] Unknown (N=101,100,98,97,97,97) | 0 | 1 | 0 | 1 | 0 | 0
  NEU [D21] Below (N=101,100,97,97,99,99) | 3 | 5 | 2 | 2 | 2 | 4
  NEU [D21] Within (N=101,100,97,97,99,99) | 97 | 92 | 91 | 93 | 92 | 88
  NEU [D21] Above (N=101,100,97,97,99,99) | 1 | 2 | 1 | 1 | 3 | 3
  NEU [D21] Unknown (N=101,100,97,97,99,99) | 0 | 1 | 3 | 1 | 2 | 4
  NEU [D28] Below (N=101,98,96,98,98,97) | 1 | 5 | 3 | 2 | 3 | 2
  NEU [D28] Within (N=101,98,96,98,98,97) | 98 | 89 | 92 | 93 | 93 | 91
  NEU [D28] Above (N=101,98,96,98,98,97) | 0 | 2 | 1 | 1 | 1 | 1
  NEU [D28] Unknown (N=101,98,96,98,98,97) | 2 | 2 | 0 | 2 | 1 | 3
  NEU [D42] Below (N=101,97,95,95,96,97) | 3 | 4 | 1 | 1 | 1 | 2
  NEU [D42] Within (N=101,97,95,95,96,97) | 98 | 91 | 94 | 92 | 93 | 93
  NEU [D42] Above (N=101,97,95,95,96,97) | 0 | 2 | 0 | 2 | 2 | 2
  NEU [D42] Unknown (N=101,97,95,95,96,97) | 0 | 0 | 0 | 0 | 0 | 0
  NEU [D63] Below (N=100,95,95,95,97,97) | 1 | 1 | 1 | 1 | 3 | 5
  NEU [D63] Within (N=100,95,95,95,97,97) | 98 | 93 | 94 | 92 | 92 | 88
  NEU [D63] Above (N=100,95,95,95,97,97) | 1 | 1 | 0 | 2 | 2 | 4
  NEU [D63] Unknown (N=100,95,95,95,97,97) | 0 | 0 | 0 | 0 | 0 | 0
  NEU [D182] Below (N=99,91,88,91,93,97) | 3 | 3 | 4 | 2 | 1 | 6
  NEU [D182] Within (N=99,91,88,91,93,97) | 93 | 86 | 83 | 86 | 89 | 89
  NEU [D182] Above (N=99,91,88,91,93,97) | 3 | 2 | 1 | 1 | 3 | 1
  NEU [D182] Unknown (N=99,91,88,91,93,97) | 0 | 0 | 0 | 2 | 0 | 1
  PLA [D0] Below (N=102,104,102,100,101,102) | 0 | 0 | 0 | 1 | 1 | 1
  PLA [D0] Within (N=102,104,102,100,101,102) | 100 | 104 | 102 | 97 | 98 | 101
  PLA [D0] Above (N=102,104,102,100,101,102) | 0 | 0 | 0 | 0 | 2 | 0
  PLA [D0] Unknown (N=102,104,102,100,101,102) | 2 | 0 | 0 | 2 | 0 | 0
  PLA [D7] Below (N=102,101,100,99,100,99) | 1 | 0 | 0 | 0 | 0 | 0
  PLA [D7] Within (N=102,101,100,99,100,99) | 101 | 100 | 100 | 97 | 99 | 99
  PLA [D7] Above (N=102,101,100,99,100,99) | 0 | 0 | 0 | 0 | 1 | 0
  PLA [D7] Unknown (N=102,101,100,99,100,99) | 0 | 1 | 0 | 2 | 0 | 0
  PLA [D21] Below (N=101,100,97,97,99,99) | 1 | 0 | 1 | 0 | 0 | 0
  PLA [D21] Within (N=101,100,97,97,99,99) | 100 | 99 | 93 | 96 | 97 | 96
  PLA [D21] Above (N=101,100,97,97,99,99) | 0 | 0 | 0 | 0 | 0 | 0
  PLA [D21] Unknown (N=101,100,97,97,99,99) | 0 | 1 | 3 | 1 | 2 | 3
  PLA [D28] Below (N=101,98,96,98,98,97) | 2 | 0 | 0 | 1 | 0 | 0
  PLA [D28] Within (N=101,98,96,98,98,97) | 98 | 96 | 96 | 96 | 95 | 94
  PLA [D28] Above (N=101,98,96,98,98,97) | 0 | 0 | 0 | 0 | 1 | 0
  PLA [D28] Unknown (N=101,98,96,98,98,97) | 1 | 2 | 0 | 1 | 2 | 3
  PLA [D42] Below (N=101,97,95,95,96,97) | 1 | 1 | 0 | 0 | 1 | 0
  PLA [D42] Within (N=101,97,95,95,96,97) | 100 | 96 | 93 | 95 | 93 | 97
  PLA [D42] Above (N=101,97,95,95,96,97) | 0 | 0 | 1 | 0 | 0 | 0
  PLA [D42] Unknown (N=101,97,95,95,96,97) | 0 | 0 | 1 | 0 | 2 | 0
  PLA [D63] Below (N=100,95,95,95,97,97) | 0 | 1 | 1 | 1 | 0 | 1
  PLA [D63] Within (N=100,95,95,95,97,97) | 100 | 94 | 94 | 93 | 96 | 96
  PLA [D63] Above (N=100,95,95,95,97,97) | 0 | 0 | 0 | 1 | 1 | 0
  PLA [D63] Unknown (N=100,95,95,95,97,97) | 0 | 0 | 0 | 0 | 0 | 0
  PLA [D182] Below (N=99,91,88,91,93,97) | 2 | 1 | 1 | 0 | 1 | 1
  PLA [D182] Within (N=99,91,88,91,93,97) | 97 | 90 | 87 | 87 | 91 | 95
  PLA [D182] Above (N=99,91,88,91,93,97) | 0 | 0 | 0 | 1 | 1 | 1
  PLA [D182] Unknown (N=99,91,88,91,93,97) | 0 | 0 | 0 | 3 | 0 | 0

15. Secondary Outcome: Microneutralization Antibody Titers Against A/California/7/2009 (H1N1) Strain.
Description: Titers were expressed as geometric mean titers (GMTs) and measured by microneutralization.
  Arepanrix vaccine strain and the unadjuvanted formulation of Arepanrix vaccine strain was A/California/7/2009 (H1N1).
  Microneutralization testing was cancelled.
Time Frame: On Days 0, 21, 42, 63 and 182
Population: Microneutralization testing was cancelled.
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Number of Subjects With a Microneutralization Titer Greater Than or Equal to 1:28 for Antibodies Against A/California/7/2009 (H1N1) Strain.
Description: Arepanrix vaccine strain and the unadjuvanted formulation of Arepanrix vaccine strain was A/California/7/2009 (H1N1).
  The antibody cut-off value assessed was a titer of 1:10 and this value was considered as seropositivity.
  Seronegative subject is a subject whose antibody titer is below the cut-off value, a seropositive subject is a subject whose antibody titer is greater than or equal to the cut-off value. Microneutralization titers < 1:28 were considered below the cut-off.
  Microneutralization testing was cancelled.
Time Frame: On Days 0, 21, 42, 63 and 182
Population: Microneutralization testing was cancelled.
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Vaccine Response Rates (VRR) for Microneutralization Antibody Titers Against A/California/7/2009 (H1N1) Strain.
Description: Arepanrix vaccine strain and the unadjuvanted formulation of Arepanrix vaccine strain was A/California/7/2009 (H1N1).
  Vaccine Response Rate for microneutralization titers was defined as the incidence rate of vaccinees with at least a 4-fold increase in post vaccination reciprocal titer relative to Day 0.
  Microneutralization testing was cancelled.
Time Frame: On Days 0, 21, 42, 63 and 182
Population: Microneutralization testing was cancelled.
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Hemagglutination Inhibition (HI) Antibody Titers Against A/California/7/2009 H1N1 Vaccine Strain.
Description: The A/California vaccine virus-homologous antibody response was measured in subjects having received two doses of Arepanrix vaccine, with prior treatment with Flulaval vaccine 21 days before the first dose and in subjects having received two doses of Arepanrix vaccine alone.
  Titers were expressed as geometric mean antibody titers (GMTs).
Time Frame: 21 days after the second dose of Arepanrix vaccine (Day 63 for Flulaval/placebo/Arepanrix Group and Day 42 for Arepanrix/placebo/Flulaval Group)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Number analyzed (Participants) | 0 | 86 | 0 | 0 | 0 | 91
Titers |  | 645.2 [557.6 to 746.6] |  |  |  | 933.1 [815.6 to 1067.6]

19. Secondary Outcome: Hemagglutination Inhibition (HI) Antibody Titers Against A/California/7/2009 H1N1 Vaccine Strain.
Description: The A/California vaccine virus-homologous antibody response was measured in subjects having received two doses of the unadjuvanted formulation of Arepanrix vaccine, with prior treatment with Flulaval vaccine 21 days before the first dose and in subjects having received two doses of the unadjuvanted formulation of Arepanrix vaccine alone.
  Titers were expressed as geometric mean antibody titers (GMTs).
Time Frame: 21 days after the second dose of the unadjuvanted formulation of Arepanrix vaccine (Day 63 for Flulaval/placebo/unadjuvanted Arepanrix Group and Day 42 for Unadjuvanted Arepanrix/placebo/Flulaval Group)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Number analyzed (Participants) | 92 | 0 | 0 | 0 | 91 | 0
Titers | 254.2 [210.1 to 307.7] |  |  |  | 387.1 [314.4 to 476.7] |

20. Secondary Outcome: Hemagglutination Inhibition (HI) Antibody Titers Against A/California/7/2009 H1N1 Vaccine Strain.
Description: The A/California vaccine virus-homologous antibody response was measured in subjects pre-treated with Flulaval who subsequently received two doses of the unadjuvanted formulation of Arepanrix vaccine compared to subjects pre-treated with Flulaval vaccine who subsequently received two doses of Arepanrix vaccine.
  Titers were expressed as geometric mean antibody titers (GMTs).
Time Frame: 21 days after the second dose of the pandemic vaccine (at Day 63)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Number analyzed (Participants) | 92 | 86 | 0 | 0 | 0 | 0
Titers | 254.2 [210.1 to 307.7] | 645.2 [557.6 to 746.6] |  |  |  |

21. Secondary Outcome: Hemagglutination Inhibition (HI) Antibody Titers Against Each of the Three Flulaval Strains.
Description: The antibody response against each of the three Flulaval vaccine components in subjects exposed to co-administration of Flulaval vaccine with the first of two doses of Arepanrix vaccine and in subjects exposed to a single dose of Flulaval vaccine.
  Flulaval vaccine strains were Flu A/Brisbane/59/2007 H1N1, Flu A/Uruguay/716/2007 H3N2 and Flu B/Brisbane/60/2008.
  Titers were expressed as geometric mean antibody titers (GMTs).
Time Frame: 21 days after the Flulaval vaccination (at Day 21).
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Number analyzed (Participants) | 92 | 86 | 0 | 89 | 0 | 0
Titers
  Flu A/BRI/59/07 H1N1 | 145.1 [115.9 to 181.6] | 215.7 [168.2 to 276.5] |  | 158.7 [127.9 to 197.1] |  |
  Flu A/Uru/716/07 H3N2 | 175.7 [129.6 to 238.2] | 183.5 [135.2 to 248.9] |  | 191.4 [138.4 to 264.7] |  |
  Flu B/Bri/60/08 | 662.1 [545.4 to 803.8] | 658.3 [540.2 to 802.0] |  | 576.1 [479.8 to 691.8] |  |

22. Secondary Outcome: Hemagglutination Inhibition (HI) Antibody Titers Against Each of the Three Flulaval Strains.
Description: The antibody response against each of the three Flulaval vaccine components in subjects exposed to co-administration of Flulaval vaccine with the first of two doses of the unadjuvanted formulation of Arepanrix vaccine and in subjects exposed to a single dose of Flulaval vaccine.
  Flulaval vaccine strains were Flu A/Brisbane/59/2007 H1N1, Flu A/Uruguay/716/2007 H3N2 and Flu B/Brisbane/60/2008.
  Titers were expressed as geometric mean antibody titers (GMTs).
Time Frame: 21 days after the Flulaval vaccination (at Day 21).
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Number analyzed (Participants) | 92 | 86 | 92 | 0 | 0 | 0
Titers
  Flu A/Brisbane/59/07 H1N1 | 145.1 [115.9 to 181.6] | 215.7 [168.2 to 276.5] | 226.3 [181.4 to 282.2] |  |  |
  Flu A/Uru/716/07 H3N2 | 175.7 [129.6 to 238.2] | 183.5 [135.2 to 248.9] | 181.7 [128.1 to 257.9] |  |  |
  Flu B/Brisbane/60/08 | 662.1 [545.4 to 803.8] | 658.3 [540.2 to 802.0] | 478.8 [389.5 to 588.6] |  |  |

23. Secondary Outcome: Hemagglutination Inhibition (HI) Antibody Titers Against Each of the Three Flulaval Strains.
Description: The antibody response against each of the three Flulaval vaccine components in subjects exposed to pre-treatment with two doses of Arepanrix vaccine and in subjects exposed to a single dose of Flulaval vaccine.
  Flulaval vaccine strains were Flu A/Brisbane/59/2007 H1N1, Flu A/Uruguay/716/2007 H3N2 and Flu B/Brisbane/60/2008.
  Titers were expressed as geometric mean antibody titers (GMTs).
Time Frame: 21 days after the Flulaval vaccination (Day 63 for Arepanrix/placebo/Flulaval Group and Day 21 for Flulaval/placebo/unadjuvanted Arepanrix and Flulaval/placebo/Arepanrix Groups)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Number analyzed (Participants) | 92 | 86 | 0 | 0 | 0 | 91
Titers
  Flu A/BRI/59/07 H1N1 | 145.1 [115.9 to 181.6] | 215.7 [168.2 to 276.5] |  |  |  | 166.9 [132.5 to 210.3]
  Flu A/Uru/716/07 H3N2 | 175.7 [129.6 to 238.2] | 183.5 [135.2 to 248.9] |  |  |  | 221.9 [167.2 to 294.6]
  Flu B/Bri/60/08 | 662.1 [545.4 to 803.8] | 658.3 [540.2 to 802.0] |  |  |  | 688.1 [593.0 to 798.6]

24. Secondary Outcome: Hemagglutination Inhibition (HI) Antibody Titers Against Each of the Three Flulaval Strains.
Description: The antibody response against each of the three Flulaval vaccine components in subjects exposed to pre-treatment with two doses of the unadjuvanted formulation of Arepanrix vaccine and in subjects exposed to a single dose of Flulaval vaccine.
  Flulaval vaccine strains were Flu A/Brisbane/59/2007 H1N1, Flu A/Uruguay/716/2007 H3N2 and Flu B/Brisbane/60/2008.
  Titers were expressed as geometric mean antibody titers (GMTs).
Time Frame: 21 days after the Flulaval vaccination (Day 63 for Unadjuvanted Arepanrix/placebo/Flulaval Group and Day 21 for Flulaval/placebo/unadjuvanted Arepanrix and Flulaval/placebo/Arepanrix Groups)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Number analyzed (Participants) | 92 | 86 | 0 | 0 | 91 | 0
Titers
  Flu A/Bri/59/07 H1N1 | 145.1 [115.9 to 181.6] | 215.7 [168.2 to 276.5] |  |  | 137.4 [109.0 to 173.1] |
  Flu A/Uru/716/07 H3N2 | 175.7 [129.6 to 238.2] | 183.5 [135.2 to 248.9] |  |  | 216.1 [160.0 to 292.0] |
  Flu B/Bri/60/08 | 662.1 [545.4 to 803.8] | 658.3 [540.2 to 802.0] |  |  | 644.9 [534.5 to 778.2] |

25. Secondary Outcome: Geometric Mean Antibody Titers (GMTs) for Hemagglutination Inhibition (HI) Antibodies Against Flu A/California H1N1 Strain.
Description: Titers were expressed as geometric mean antibody titers (GMTs).
Time Frame: On Days 0, 21, 42 and 63
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Number analyzed (Participants) | 92 | 86 | 92 | 89 | 91 | 91
Titers
  Flu A/Cal H1N1 [at Day 0] (N=92;86;92;88;91;91) | 14.6 [11.2 to 19.0] | 10.9 [8.7 to 13.6] | 13.0 [10.2 to 16.5] | 10.7 [8.2 to 14.0] | 9.3 [7.7 to 11.4] | 10.1 [8.2 to 12.5]
  Flu A/Cal H1N1 [at Day 21] (N=92;86;92;89;91;91) | 31.1 [24.0 to 40.3] | 26.3 [19.9 to 34.8] | 277.3 [222.4 to 345.7] | 361.0 [301.5 to 432.2] | 358.7 [285.0 to 451.4] | 659.8 [546.0 to 797.4]
  Flu A/Cal H1N1 [at Day 42] (N=92;86;92;89;91;91) | 238.6 [191.8 to 296.7] | 396.2 [329.2 to 476.8] | 271.2 [224.6 to 327.4] | 589.8 [517.8 to 671.8] | 387.1 [314.4 to 476.7] | 933.1 [815.6 to 1067.6]
  Flu A/Cal H1N1 [at Day 63] (N=92;86;92;89;91;91) | 254.2 [210.1 to 307.7] | 645.2 [557.6 to 746.6] | 245.0 [200.7 to 299.1] | 426.9 [373.0 to 488.5] | 345.3 [278.6 to 428.0] | 704.0 [602.1 to 823.1]

26. Secondary Outcome: Geometric Mean Antibody Titers (GMTs) for Hemagglutination Inhibition (HI) Antibodies Against Flu A/California H1N1 Strain.
Description: Titers were expressed as geometric mean antibody titers (GMTs).
Time Frame: At Day 182
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Number analyzed (Participants) | 92 | 89 | 85 | 89 | 89 | 91
Titers | 136.6 [108.6 to 171.9] | 206.9 [171.3 to 249.9] | 151.7 [119.1 to 193.2] | 171.7 [143.2 to 205.8] | 218.5 [169.8 to 281.1] | 323.6 [268.8 to 389.5]

27. Secondary Outcome: Number of Seroconverted Subjects for Antibodies Against A/ California Strain.
Description: Seroconversion rate was defined as the incidence rate of vaccinees who had either a pre-vaccination titer recorded as < 1:10 and a post-vaccination reciprocal titer ≥ 40 or a pre-vaccination reciprocal titer ≥ 10 and at least a 4-fold increase in post vaccination reciprocal titer.
  Seroconversion defined as:
  For initially seronegative subjects, antibody titer ≥ 1:40 after vaccination For initially seropositive subjects, antibody titer after vaccination ≥ 4 fold the pre-vaccination antibody titer
Time Frame: At Day 63 from Day 21 for Flulaval/placebo/unadjuvanted Arepanrix and Flulaval/placebo/Arepanrix Groups; At Day 42 from Day 0 for the 4 other groups
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Number analyzed (Participants) | 92 | 86 | 92 | 88 | 91 | 91
Subjects | 66 | 77 | 84 | 85 | 88 | 90

28. Secondary Outcome: Number of Seroprotected Subjects for Antibodies Against A/California Strain.
Description: Seroprotection rate was defined as the proportion of subjects with H1N1 reciprocal HI titers ≥ 40 against the tested vaccine virus.
Time Frame: At Day 63 for Flulaval/placebo/unadjuvanted Arepanrix and Flulaval/placebo/Arepanrix Groups; At Day 42 for the 4 other groups.
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Number analyzed (Participants) | 92 | 86 | 92 | 89 | 91 | 91
Subjects | 90 | 86 | 92 | 89 | 91 | 91

29. Secondary Outcome: Seroconversion Factor for Antibodies Against A/California Strain.
Description: Seroconversion factor was defined as the geometric mean of the within-subject ratios of the post-vaccination reciprocal HI titer to the prevaccination reciprocal HI titer.
Time Frame: as for outcome 27
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Fold
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Number analyzed (Participants) | 92 | 86 | 92 | 88 | 91 | 91
Fold | 8.2 [6.4 to 10.5] | 24.6 [18.1 to 33.3] | 20.9 [16.3 to 26.7] | 54.9 [42.1 to 71.7] | 41.5 [32.4 to 53.2] | 92.4 [73.3 to 116.3]

30. Secondary Outcome: Number of Seroconverted Subjects for Antibodies Against Flulaval Vaccine Strains.
Description: Seroconversion defined as:
  For initially seronegative subjects, antibody titer ≥ 1:40 after vaccination For initially seropositive subjects, antibody titer after vaccination ≥ 4 fold the pre-vaccination antibody titer
  Flulaval vaccines strains were A/Brisbane/59/2007 H1N1, A/Uruguay/716/2007 H3N2 and B/Brisbane/60/2008.
  For the analysis the Flulaval/placebo/unadjuvanted Arepanrix Group and the Flulaval/placebo/Arepanrix Group were pooled.
Time Frame: At Day 21 from Day 0 for the pooled group, Flulaval/unadjuvanted Arepanrix/placebo and Flulaval/Arepanrix/placebo Groups; at Day 63 from Day 42 for Unadjuvanted Arepanrix/placebo/Flulaval Group and Arepanrix/placebo/Flulaval Group
Population: as for outcome 1
Measure: Number; unit: Subjects
Groups:
- Flulaval/Placebo/(Unadjuvanted) Arepanrix Pooled Group: subjects received co-administration of Flulaval vaccine and saline placebo on Day 0 followed by the (unadjuvanted formulation of ) Arepanrix vaccine on Day 21 and Day 42. All vaccines were administered intramuscularly in the deltoids of the dominant or non dominant arm. At Day 0 the two vaccines were administered each in a separate arm, at Day 21 in the dominant arm and at Day 42 in the non-dominant arm.
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group | Flulaval/Placebo/(Unadjuvanted) Arepanrix Pooled Group
Number analyzed (Participants) | 0 | 0 | 92 | 88 | 91 | 91 | 178
Subjects
  Flu A/Bri/59/07 H1N1 |  |  | 76 | 70 | 50 | 33 | 145
  Flu A/Uru/716/07 H3N2 |  |  | 72 | 76 | 73 | 72 | 145
  Flu B/Bri/60/08 |  |  | 74 | 78 | 71 | 57 | 152

31. Secondary Outcome: Number of Seroprotected Subjects for Antibodies Against Flulaval Vaccine Strains
Description: Seroprotection was defined as the proportion of subjects with H1N1 reciprocal Hemagglutination Inhibition (HI) titers ≥ 1:40 against the tested vaccine virus.
  Flulaval vaccines strains were A/Brisbane/59/2007 H1N1, A/Uruguay/716/2007 H3N2 and B/Brisbane/60/2008.
  For the analysis the Flulaval/placebo/unadjuvanted Arepanrix Group and the Flulaval/placebo/Arepanrix Group were pooled.
Time Frame: At Day 21 for the pooled group, Flulaval/unadjuvanted Arepanrix/placebo and Flulaval/Arepanrix/placebo Groups; at Day 63 for Unadjuvanted Arepanrix/placebo/Flulaval Group and Arepanrix/placebo/Flulaval Group
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group | Flulaval/Placebo/(Unadjuvanted) Arepanrix Pooled Group
Number analyzed (Participants) | 0 | 0 | 92 | 89 | 91 | 91 | 178
Subjects
  Flu A/Bri/59/07 H1N1 |  |  | 89 | 82 | 81 | 87 | 170
  Flu A/Uru/716/07 H3N2 |  |  | 77 | 79 | 81 | 83 | 155
  Flu B/Bri/60/08 |  |  | 90 | 89 | 91 | 91 | 176

32. Secondary Outcome: Seroconversion Factor for Antibodies Against Flulaval Vaccine Strains.
Description: Seroconversion factor was defined as the geometric mean of the within-subject ratios of the post-vaccination reciprocal Hemagglutination Inhibition (HI) titer to the prevaccination reciprocal HI titer.
  Flulaval vaccines strains were A/Brisbane/59/2007 H1N1, A/Uruguay/716/2007 H3N2 and B/Brisbane/60/2008.
  For the analysis the Flulaval/placebo/unadjuvanted Arepanrix Group and the Flulaval/placebo/Arepanrix Group were pooled.
Time Frame: as for outcome 30
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Fold
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group | Flulaval/Placebo/(Unadjuvanted) Arepanrix Pooled Group
Number analyzed (Participants) | 0 | 0 | 92 | 88 | 91 | 91 | 178
Fold
  Flu A/Bri/59/07 H1N1 |  |  | 12.0 [9.4 to 15.4] | 9.6 [7.7 to 12.1] | 4.2 [3.5 to 5.0] | 3.1 [2.5 to 3.9] | 10.3 [8.6 to 12.3]
  Flu A/Uru/716/07 H3N2 |  |  | 20.6 [14.8 to 28.6] | 19.3 [14.2 to 26.4] | 17.3 [12.8 to 23.2] | 11.6 [8.9 to 15.2] | 16.5 [13.5 to 20.1]
  Flu B/Bri/60/08 |  |  | 10.5 [8.3 to 13.5] | 14.3 [11.0 to 18.7] | 8.6 [7.0 to 10.7] | 4.9 [4.1 to 6.0] | 13.2 [11.1 to 15.7]

33. Secondary Outcome: Number of Seroconverted Subjects for Antibodies Against Flulaval Vaccine Strains
Description: Seroconversion defined as:
  For initially seronegative subjects, antibody titer ≥ 1:40 after vaccination For initially seropositive subjects, antibody titer after vaccination ≥ 4 fold the pre-vaccination antibody titer
  Flulaval vaccines strains were A/Brisbane/59/2007 H1N1, A/Uruguay/716/2007 H3N2 and B/Brisbane/60/2008.
Time Frame: on Days 21 and 63 from Day 0 for the first 4 groups; on Days 42 and 63 from Day 0 for the Unadjuvanted Arepanrix/placebo/Flulaval and Arepanrix/placebo/Flulaval Groups
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Number analyzed (Participants) | 92 | 86 | 92 | 88 | 91 | 91
Subjects
  Flu A/Bri/59/07 H1N1 [Day 21 or 42 after dose 1] | 71 | 74 | 76 | 70 | 17 | 28
  Flu A/Bri/59/07 H1N1 [Day 63 after dose 1] | 63 | 76 | 69 | 64 | 71 | 76
  Flu A/Uru/716/07 H3N2 [Day 21 or 42 after dose 1] | 72 | 73 | 72 | 76 | 3 | 6
  Flu A/Uru/716/07 H3N2 [Day 63 after dose 1] | 71 | 69 | 69 | 69 | 75 | 78
  Flu B/Bri/60/08 [Day 21 or 42 after dose 1] | 76 | 76 | 74 | 78 | 6 | 24
  Flu B/Bri/60/08 [Day 63 after dose 1] | 73 | 73 | 67 | 73 | 78 | 76

34. Secondary Outcome: Number of Seroconverted Subjects for Antibodies Against Flulaval Vaccine Strains
Description: as for outcome 33
Time Frame: At Day 182 from Day 0
Population: as for outcome 3
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Number analyzed (Participants) | 92 | 89 | 85 | 88 | 89 | 91
Subjects
  Flu A/Bri/59/07 H1N1 | 45 | 57 | 45 | 38 | 46 | 54
  Flu A/Uru/716/07 H3N2 | 58 | 56 | 54 | 56 | 60 | 61
  Flu B/Bri/60/08 Victoria | 68 | 54 | 48 | 64 | 67 | 62

35. Secondary Outcome: Number of Seroprotected Subjects for Antibodies Against Flulaval Vaccine Strains.
Description: Seroprotection rate was defined as the proportion of subjects with H1N1 reciprocal HI titers ≥ 40 against the tested vaccine virus.
  Flulaval vaccines strains were A/Brisbane/59/2007 H1N1, A/Uruguay/716/2007 H3N2 and B/Brisbane/60/2008.
Time Frame: before vaccination and on days 21 and 63 for the first 4 groups and before vaccination and on days 42 and 63 for the Unadjuvanted Arepanrix/placebo/Flulaval and Arepanrix/placebo/Flulaval Groups
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Number analyzed (Participants) | 92 | 86 | 92 | 89 | 91 | 91
Subjects
  Flu A/Bri/59/07 H1N1 [at Day 0] | 20 | 18 | 26 | 18 | 23 | 20
  Flu A/Bri/59/07 H1N1 [Days 21 or 42 post dose 1] | 86 | 84 | 89 | 82 | 47 | 62
  Flu A/Bri/59/07 H1N1 [at Day 63 post dose 1] | 84 | 86 | 85 | 79 | 81 | 87
  Flu A/Uru/716/07 H3N2 [at Day 0] | 12 | 16 | 8 | 13 | 15 | 17
  Flu A/Uru/716/07 H3N2 [Days 21 or 42 post dose 1] | 78 | 77 | 77 | 79 | 18 | 28
  Flu A/Uru/716/07 H3N2 [at Day 63 post dose 1] | 78 | 75 | 73 | 75 | 81 | 83
  Flu B/Bri/60/08 [at Day 0] | 62 | 50 | 56 | 49 | 66 | 62
  Flu B/Bri/60/08 [Days 21 or 42 post dose 1] | 91 | 85 | 90 | 89 | 75 | 89
  Flu B/Bri/60/08 [at Day 63 post dose 1] | 91 | 86 | 91 | 89 | 91 | 91

36. Secondary Outcome: Number of Seroprotected Subjects for Antibodies Against Flulaval Vaccine Strains.
Description: as for outcome 35
Time Frame: At Day 182 after the first dose
Population: as for outcome 3
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Number analyzed (Participants) | 92 | 89 | 85 | 89 | 89 | 91
Subjects
  Flu A/Bri/59/07 H1N1 | 63 | 74 | 66 | 61 | 67 | 71
  Flu A/Uru/716/07 H3N2 | 66 | 64 | 60 | 64 | 68 | 70
  Flu B/Bri/60/08 Victoria | 90 | 88 | 79 | 89 | 88 | 91

37. Secondary Outcome: Seroconversion Factor for Antibodies Against Flulaval Vaccine Strains.
Description: Seroconversion factor of the within-subject ratios of the post-vaccination reciprocal HI titer to the Day 0 reciprocal HI titer.
  Flulaval vaccines strains were A/Brisbane/59/2007 H1N1, A/Uruguay/716/2007 H3N2 and B/Brisbane/60/2008.
Time Frame: On Days 21 and 63 from Day 0 for the first 4 groups and on Days 42 and 63 from Day 0 for the Unadjuvanted Arepanrix/placebo/Flulaval and Arepanrix/placebo/Flulaval Groups
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Fold
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Number analyzed (Participants) | 92 | 86 | 92 | 88 | 91 | 91
Fold
  Flu A/Bri/59/07 H1N1 [Day 21 or 42 post dose 1] | 8.4 [6.5 to 10.8] | 12.9 [10.0 to 16.6] | 12.0 [9.4 to 15.4] | 9.6 [7.7 to 12.1] | 2.3 [1.9 to 2.6] | 3.2 [2.7 to 3.8]
  Flu A/Bri/59/07 H1N1 [at Day 63 post dose 1] | 6.9 [5.4 to 8.9] | 11.2 [9.1 to 13.7] | 8.4 [6.6 to 10.6] | 7.6 [6.0 to 9.5] | 9.4 [7.6 to 11.7] | 10.1 [8.1 to 12.6]
  Flu A/Uru/716/07 H3N2 [Day 21 or 42 post dose 1] | 17.4 [13.0 to 23.3] | 15.5 [11.8 to 20.4] | 20.6 [14.8 to 28.6] | 19.3 [14.2 to 26.4] | 1.2 [1.1 to 1.4] | 1.7 [1.5 to 1.9]
  Flu A/Uru/716/07 H3N2 [at Day 63 post dose 1] | 13.3 [10.0 to 17.6] | 11.7 [9.1 to 15.0] | 15.0 [11.2 to 19.9] | 14.6 [10.9 to 19.6] | 20.8 [15.5 to 28.0] | 19.3 [14.6 to 25.5]
  Flu B:Bri/60/08 [Day 21 or 42 post dose 1] | 12.6 [9.8 to 16.2] | 13.9 [11.1 to 17.5] | 10.5 [8.3 to 13.5] | 14.3 [11.0 to 18.7] | 1.3 [1.1 to 1.5] | 2.4 [2.0 to 2.8]
  Flu B/Bri/60/08 [at Day 63 post dose 1] | 9.6 [7.5 to 12.4] | 10.0 [8.1 to 12.2] | 7.9 [6.3 to 9.9] | 10.8 [8.4 to 13.7] | 11.4 [9.1 to 14.2] | 11.9 [9.4 to 15.0]

38. Secondary Outcome: Seroconversion Factor for Antibodies Against Flulaval Vaccine Strains.
Description: as for outcome 37
Time Frame: At Day 182 from Day 0
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: Fold
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Number analyzed (Participants) | 92 | 89 | 85 | 88 | 89 | 91
Fold
  Flu A/Bri/59/07 H1N1 | 4.0 [3.1 to 5.3] | 5.2 [4.2 to 6.6] | 4.7 [3.7 to 6.0] | 3.7 [2.9 to 4.8] | 4.4 [3.5 to 5.4] | 5.0 [4.0 to 6.3]
  Flu A/Uru/716/07 H3N2 | 9.0 [6.7 to 11.9] | 7.2 [5.6 to 9.3] | 9.7 [7.2 to 13.1] | 8.5 [6.2 to 11.7] | 9.9 [7.3 to 13.5] | 10.6 [7.9 to 14.2]
  Flu B/Bri/60/08 Victoria | 6.7 [5.2 to 8.6] | 5.7 [4.5 to 7.1] | 5.5 [4.3 to 6.9] | 6.8 [5.3 to 8.6] | 6.9 [5.4 to 8.7] | 6.4 [5.0 to 8.1]

39. Secondary Outcome: Geometric Mean Antibody Titers (GMTs) for Hemagglutination Inhibition (HI) Antibodies Against Flulaval Vaccine Strains.
Description: Titers were expressed as geometric mean titers (GMTs).
  Flulaval vaccines strains were A/Brisbane/59/2007 H1N1, A/Uruguay/716/2007 H3N2 and B/Brisbane/60/2008.
Time Frame: On Days 0, 21 and 63 for the first 4 groups and on Days 0, 42 and 63 for the Unadjuvanted Arepanrix/placebo/Flulaval and Arepanrix/placebo/Flulaval Groups
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Number analyzed (Participants) | 92 | 86 | 92 | 89 | 91 | 91
Titers
  Flu A/Bri/59/07 H1N1 [at Day 0] | 17.3 [14.1 to 21.3] | 16.7 [13.8 to 20.2] | 18.8 [15.2 to 23.3] | 16.2 [12.8 to 20.6] | 14.6 [12.0 to 17.8] | 16.6 [13.7 to 20.0]
  Flu A/Bri/59/07 H1N1 [at Day 21 or 42] | 145.1 [115.9 to 181.6] | 215.7 [168.2 to 276.5] | 226.3 [181.4 to 282.2] | 158.7 [127.9 to 197.1] | 32.9 [27.3 to 39.7] | 53.2 [43.5 to 65.1]
  Flu A/Bri/59/07 H1N1 [at Day 63] | 120.2 [96.5 to 149.7] | 186.5 [150.4 to 231.4] | 157.0 [126.0 to 195.8] | 124.3 [99.0 to 156.1] | 137.4 [109.0 to 173.1] | 166.9 [132.5 to 210.3]
  Flu A/Uru/716/07 H3N2 [at Day 0] | 10.1 [8.1 to 12.5] | 11.8 [9.7 to 14.4] | 8.8 [7.4 to 10.6] | 10.2 [8.3 to 12.6] | 10.4 [8.4 to 12.8] | 11.5 [9.4 to 14.1]
  Flu A/Uru/716/07 H3N2 [at Day 21 or 42] | 175.7 [129.6 to 238.2] | 183.5 [135.2 to 248.9] | 181.7 [128.1 to 257.9] | 191.4 [138.4 to 264.7] | 12.5 [10.0 to 15.6] | 19.1 [15.6 to 23.4]
  Flu A/Uru/716/07 H3N2 [at Day 63] | 134.4 [100.4 to 179.9] | 138.4 [104.8 to 182.7] | 132.0 [94.9 to 183.7] | 145.6 [107.7 to 196.8] | 216.1 [160.0 to 292.0] | 221.9 [167.2 to 294.6]
  Flu B/Bri/60/08 [at Day 0] | 52.6 [41.8 to 66.3] | 47.3 [38.0 to 58.9] | 45.4 [36.0 to 57.4] | 40.1 [31.5 to 51.1] | 56.7 [45.7 to 70.5] | 58.0 [47.2 to 71.4]
  Flu B/Bri/60/08 [at Day 21 or 42] | 662.1 [545.4 to 803.8] | 658.3 [540.2 to 802.0] | 478.8 [389.5 to 588.6] | 576.1 [479.8 to 691.8] | 74.7 [61.4 to 90.9] | 139.5 [120.0 to 162.2]
  Flu B/Bri/60/08 [at Day 63] | 506.7 [422.3 to 608.0] | 471.2 [396.3 to 560.2] | 359.6 [299.4 to 431.9] | 433.5 [369.5 to 508.7] | 644.9 [534.5 to 778.2] | 688.1 [593.0 to 798.6]

40. Secondary Outcome: Geometric Mean Antibody Titers (GMTs) for Hemagglutination Inhibition (HI) Antibodies Against Flulaval Vaccine Strains.
Description: as for outcome 39
Time Frame: At Day 182 after dose 1 vaccination
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Number analyzed (Participants) | 92 | 89 | 85 | 89 | 89 | 91
Titers
  Flu A/Bri/59/07 H1N1 | 68.5 [53.6 to 87.4] | 89.2 [71.0 to 112.0] | 87.4 [68.5 to 111.5] | 64.6 [51.4 to 81.1] | 64.6 [51.4 to 81.1] | 83.7 [66.0 to 106.2]
  Flu A/Uru/716/07 H3N2 | 89.5 [65.8 to 121.8] | 87.7 [64.0 to 120.3] | 87.1 [61.4 to 123.5] | 87.8 [63.4 to 121.4] | 110.0 [79.3 to 152.6] | 127.2 [92.3 to 175.5]
  Flu B/Bri/60/08 Victoria | 339.9 [276.7 to 417.5] | 273.8 [228.7 to 327.9] | 245.4 [197.8 to 304.3] | 292.6 [247.0 to 346.7] | 369.6 [300.0 to 455.3] | 378.4 [323.4 to 442.8]

ADVERSE EVENTS:
Time Frame: SAEs:during the entire study period (Days 0-329). Unsolicited AEs: within the 84-day (Days 0-83) post-vaccination period. Solicited symptoms: During a 7-day follow-up period (Days 0-6) after vaccination
Description: SAEs were collected up to Day 329 which corresponds to the last contact day with the subjects reporting serious adverse events.
Arm/Group | Flulaval/Placebo/Unadjuvanted Arepanrix Group | Flulaval/Placebo/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix/Placebo Group | Flulaval/Arepanrix/Placebo Group | Unadjuvanted Arepanrix/Placebo/Flulaval Group | Arepanrix/Placebo/Flulaval Group
Serious Adverse Events (participants affected / at risk) | 3/102 | 1/104 | 1/102 | 2/100 | 1/101 | 3/102
Other Adverse Events (participants affected / at risk) | 92/102 | 91/104 | 86/102 | 97/100 | 84/101 | 99/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Flulaval/Placebo/Unadjuvanted Arepanrix Group (N=102) | Flulaval/Placebo/Arepanrix Group (N=104) | Flulaval/Unadjuvanted Arepanrix/Placebo Group (N=102) | Flulaval/Arepanrix/Placebo Group (N=100) | Unadjuvanted Arepanrix/Placebo/Flulaval Group (N=101) | Arepanrix/Placebo/Flulaval Group (N=102)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Flulaval/Placebo/Unadjuvanted Arepanrix Group (N=102) | Flulaval/Placebo/Arepanrix Group (N=104) | Flulaval/Unadjuvanted Arepanrix/Placebo Group (N=102) | Flulaval/Arepanrix/Placebo Group (N=100) | Unadjuvanted Arepanrix/Placebo/Flulaval Group (N=101) | Arepanrix/Placebo/Flulaval Group (N=102)
Upper respiratory tract infection (Infections and infestations) | 11 | 11 | 11 | 8 | 15 | 11
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 | 17 | 9 | 12 | 6 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 11 | 11 | 6 | 11 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 | 7 | 0 | 0 | 8 | 5
Nasopharyngitis (Infections and infestations) | 0 | 0 | 10 | 0 | 7 | 0
Nausea (Gastrointestinal disorders) | 9 | 8 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 7 | 0 | 6 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 7 | 6 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 8
Pain (General disorders) | 75 | 89/100 | 66/100 | 94/99 | 69 | 95/100
Redness (General disorders) | 2 | 6/100 | 1/100 | 5/99 | 1 | 11/100
Swelling (General disorders) | 2 | 15/100 | 2/100 | 9/99 | 0 | 16/100
Fatigue (General disorders) | 54 | 62/100 | 41/100 | 58/99 | 57 | 56/100
Headache (General disorders) | 52 | 58/100 | 51/100 | 51/99 | 49 | 54/100
Joint pain at other location (General disorders) | 24 | 34/100 | 24/100 | 28/99 | 26 | 23/100
Muscle aches (General disorders) | 38 | 52/100 | 39/100 | 53/99 | 43 | 54/100
Shivering (General disorders) | 21 | 30/100 | 19/100 | 24/99 | 21 | 25/100
Sweating (General disorders) | 22 | 21/100 | 21/100 | 17/99 | 12 | 25/100
Temperature (General disorders) | 3 | 9/100 | 3/100 | 2/99 | 1 | 4/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.